



# **ITC 6 European Country Survey**

**Wave 1 Technical Report** 

**February 1, 2017** 



This project has received funding from the European Union's Horizon 2020 research and innovation programme under grant agreement No 681109

### ITC 6 European Country Research Team

Dr. Constantine Vardavas<sup>1</sup>, Principal Investigator and EUREST-PLUS Coordinator

Dr. Ute Mons<sup>2</sup>, Principal Investigator, Germany

Dr. Yannis Tountas<sup>3</sup>, Principal Investigator, Greece

Mr. Tibor Demjén<sup>4</sup>, Principal Investigator, Hungary

Mr. Krzysztof Przewoźniak<sup>5</sup>, Principal Investigator, Poland

Dr. Witold Zatoński<sup>5</sup>, Principal Investigator, Poland

Dr. Antigona Trofor<sup>6</sup>, Principal Investigator, Romania

Dr. Esteve Fernandez<sup>7</sup>, Principal Investigator, Spain

Mr. Nicolas Bécuwe<sup>8</sup>, Principal Investigator, Belgium

Ms. Sophie Goudet<sup>8</sup>, Co-investigator, Belgium

Mr. Christopher Hanley<sup>8</sup>, Data Analyst. Belgium

ITC 6 European Country International Research Team Professor Geoffrey T. Fong<sup>9</sup>, Principal Investigator, Canada

Professor Mary E. Thompson<sup>10</sup>, Co-Investigator, Canada

Dr. Shannon Gravely<sup>9</sup>, Co-Investigator, Canada

Dr. Anne C.K. Quah<sup>9</sup>, Co-investigator, Canada

Mr. Thomas Agar<sup>9</sup>, Project Manager, Canada

Mr. Pete Driezen<sup>9</sup>, Senior Data Analyst, Canada

**Funding:** The ITC 6 European Country Project has received funding support from:

- European Union's Horizon 2020 Program (Grant No. 681109 Vardavas)
- University of Waterloo, Canada (Grant No. 118096 Fong)

Suggested Citation: ITC Project. (2017, January). ITC 6 European Country Wave 1 (2016) Technical Report. University of Waterloo, Waterloo, Ontario, Canada, and European Network on Smoking and Tobacco Prevention, Brussels, Belgium.

<sup>&</sup>lt;sup>1</sup> European Network on Smoking and Tobacco Prevention

<sup>&</sup>lt;sup>2</sup> German Cancer Research Center

<sup>&</sup>lt;sup>3</sup>University of Athens, Medical School

<sup>&</sup>lt;sup>4</sup> Smoking or Health Hungarian Foundation (SHHF)

<sup>&</sup>lt;sup>5</sup> Health Promotion Foundation

<sup>&</sup>lt;sup>6</sup> Aer Pur Romania

<sup>&</sup>lt;sup>7</sup> Institut CatalÃă dâĂŹOncologia

<sup>&</sup>lt;sup>8</sup> Kantar Public

<sup>&</sup>lt;sup>9</sup> Department of Psychology, University of Waterloo

<sup>&</sup>lt;sup>10</sup> Department of Statistics and Actuarial Science, University of Waterloo

# **Contents**

| Pı | eface | e | 5 |
|----|-------|-------------------------------------------------------|----|
| 1 | Intr | roduction | 6 |
| | 1.1 | Background | 6 |
| | 1.2 | Main Objectives | 7 |
| | 1.3 | Survey Design | 9 |
| | 1.4 | The Research Team | 9 |
| | 1.5 | Country Timelines | 10 |
| 2 | Sur | vey Process, Protocols and Fieldwork | 23 |
| | 2.1 | Survey Process | 23 |
| | 2.2 | Replenishment Participant Selection and Consent | 23 |
| | 2.3 | Household Screener Survey | 24 |
| | 2.4 | Main Questionnaire | 24 |
| | | 2.4.1 Screeners | 24 |
| | | 2.4.2 Content of Survey | 25 |
| | | 2.4.3 Language of Survey | 25 |
| | | 2.4.4 Length of the Interview | 25 |
| | 2.5 | Remuneration | 25 |
| | 2.6 | Progress Report | 26 |
| | | 2.6.1 Survey Translation | 26 |
| | | 2.6.2 Field Work Preparation and Interviewer Training | 26 |
| | | 2.6.3 Survey Fieldwork | 26 |
| | | 2.6.4 Questionnaire Checking | 27 |
| | | 2.6.5 Data Checking and Cleaning | 28 |
| | | 2.6.6 Data Delivery | 28 |

# CONTENTS

| 3 | Mor | nitoring and Quality Control | <b>29</b> |
|----|------|-----------------------------------------------------|-----------|
| | 3.1 | Management of Fieldwork Teams | 29 |
| | 3.2 | Survey Protocol | 29 |
| | 3.3 | Monitoring and Quality Assurance | 29 |
| | 3.4 | Handling Special Situations | 30 |
| 4 | Sam | pling Design and Weight Construction | 31 |
| | 4.1 | Sampling design | 31 |
| | 4.2 | Weight construction | 32 |
| | | 4.2.1 General comments about weight construction | 32 |
| | | 4.2.2 Wave 1 weights | 33 |
| | 4.3 | Taking the sampling design into account in analyses | 36 |
| | | 4.3.1 Specification of strata and PSUs for analyses | 36 |
| | | 4.3.2 Bootstrap weights | 37 |
| Ap | pen | dices | <b>39</b> |
| A | Sam | aple size tables | <b>39</b> |
| В | Ben | chmark/calibration figures | <b>39</b> |
| C | Sun | nmary statistics of the weights | <b>58</b> |
| D | Fiel | d materials | 63 |
| E | Sur | vey information letter and consent | 63 |
| F | Fina | al outcomes rates | <b>67</b> |
| G | Cou | intry profiles | <b>69</b> |

# **Preface**

This technical report documents the first wave of the International Tobacco Control Policy Evaluation Survey carried out in Germany, Greece, Hungary, Poland, Romania, and Spain. This project is known as the ITC 6 European Country Project (6E) under the larger project called European Regulatory Science on Tobacco: Policy Implementation to Reduce Lung Disease (EUREST-PLUS). Wave 1 was conducted from June to September 2016.

This report also presents the weight calculations for the Wave 1 respondents.

# 1 Introduction

# 1.1 Background

The International Tobacco Control (ITC) Project is a multi-country prospective cohort study designed to measure the psychosocial and behavioural impact of key policies of the World Health Organization (WHO) Framework Convention on Tobacco Control (FCTC).

Germany, Greece, Hungary, Poland, Romania, and Spain make up the six countries of the ITC 6 European Country Project (6E). Hungary was the first state to ratify the FCTC in April 2004, followed by Germany in December of that year. Spain ratified the FCTC in January 2005. Greece was next to ratify the FCTC in January 2006, followed by the remaining states (Poland and Romania) in September 2006. In addition to the FCTC, each country is a party of the European Union, and as such must also comply with the European Commission's Tobacco Products Directive (TPD), the latest of which was made law in 2014 with a compliance date of May 20, 2016. Previous to the TPD of 2014 was the TPD of 2001, under which all six European States had to meet minimum standards of tobacco labelling and packaging restrictions, as well as regulations regarding cross-border trading and product ingredients. The latest TPD (2014) sets regulations on the following areas:

- (i) Ingredients and emissions, including maximum emission levels on tar, nicotine, and CO<sub>2</sub>, as well as restrictions on additives such as flavours and stimulants
- (ii) Labelling and packaging restrictions, setting minimum dimensions for packages of tobacco as minimum standards on graphic (combined) tobacco health warning labels
- (iii) Traceability and security measures to combat illegal cigarette smuggling and counterfeit products
- (iv) Cross-border purchase regulations
- (v) E-cigarette product regulations including pan-European restrictions on the amount of nicotine allowed within e-cigarettes/e-liquid, product design elements such as reservoir sizes, and more.

To evaluate the effect of the FCTC and the TPD (2014), the ITC Project is conducting the ITC 6E Project as part of the European Regulatory Science on Tobacco: Policy Implementation to Reduce Lung Disease (EUREST PLUS) Project. The main objective of EUREST-PLUS Project is to monitor and evaluate the impact of the implementing acts of the TPD and assess these within the context of FCTC ratification at a European level.

The ITC 6E Project will run two prospective cohort surveys which will parallel surveys of adult smokers in 22 other ITC countries—(Canada, United States, United Kingdom, Australia, Ireland, Thailand, Malaysia, China, South Korea, New Zealand, Mexico, Uruguay, France, The Netherlands, Brazil, Mauritius, Bangladesh, Bhutan, India, Kenya, Zambia, and Abu Dhabi – United Arab Emirates).

The ITC 6 European Country Wave 1 Survey was carried out from June to September 2016.

# **Main Objectives**

Representing three of the seven work packages (WP) of the EUREST-PLUS Project, the ITC 6 European Country Project is key to meeting the overall EUREST-PLUS objectives. Those objectives are:

- a) To evaluate the psychosocial and behavioral impact of TPD implementation and FCTC implementation, through the creation of a longitudinal cohort of adult smokers in 6 EU MS (Germany, Greece, Hungary, Poland, Romania, and Spain; total n=6000) in a pre- vs. post-TPD study design (Work Package, or WP, 2 and 3). Moreover, these evaluation studies of the impact of the TPD and FCTC will be conducted with respect to vulnerable populations, including low-income/socio-economic status (SES) groups and those smokers with respiratory co-morbidities (and/or those with pre-morbid symptomatology). Another important topic that will be addressed in the scientific studies of the ITC 6E cohorts will be a focus on e-cigarettes, addressing basic issues of transition rates from cigarettes to e-cigarettes or dual use, rates of reversion back to cigarettes and rates of quitting all nicotine products. Studies that examine e-cigarettes will be linked to additional analysis, focussing on product testing of various design features of e-cigarettes systematically procured in those same 6 countries where the ITC 6 European Country Surveys will be conducted.
- b) To assess support for TPD implementation through secondary dataset analyses of the 2015 Special Eurobarometer on Tobacco Survey (SETS), a cross-sectional survey performed among 27,000 adults in all 28 EU MS, before the TPD is implemented, and to monitor progress in FCTC implementation in the EU over the past years through trend analyses on the merged datasets of the 2009, 2012 and 2015 SETS datasets (n=80,000), with a special focus on vulnerable populations (youth, minorities, unemployed, etc.) (WP5)
- c) To document changes in e-cigarette product parameters (technical design, labelling/ packaging and chemical composition) following TPD implementation of Article 20 of the TPD. (WP6)
- d) To enhance innovative joint research collaborations on chronic, non-communicable diseases (NCDs) in low- and middle-income countries (LMICs) and in vulnerable populations in high-income countries (HICs), a key priority of the Global Alliance for Chronic Disease (GACD) outlined in the call. We will specifically address these crosscountry analyses through the pooling and comparisons across both other EU countries of the ITC Project (6E, UK, France, Netherlands), and other non-EU countries from LMICs and HICs from the global ITC Project (including key countries of comparison such as Australia, Canada, New Zealand, United States, China). (WP4)

The objectives of the ITC 6 European Country Survey are:

- a. To examine the prevalence and patterns of tobacco use in all six European States. The ITC 6 European Country Survey provides multidimensional estimates of prevalence and patterns of tobacco use among the populations of all six participating states. It describes the consumption patterns and quitting behaviour within each country's population, as well as each population's knowledge, beliefs, and attitudes about tobacco use. As well, the survey investigates each country's growth or absence of awareness and use of electronic cigarettes (e-cigarettes).
- b. To examine the impact of the Tobacco Products Directive (2014) in all 6 countries throughout the course of the study period. The ITC 6E Survey evaluates the impact of the TPD in the following areas:
  - Health warning labels and package descriptors
  - Tobacco ingredients and additives
  - Cross-border sales of tobacco products
  - · E-cigarette use and behaviour

The survey also evaluates the impact of the FCTC in the following areas:

- Smoke-free legislation
- Pricing and taxation of tobacco products, as well as the prevalence of compensatory behaviours that may offset the impact of taxation (e.g., cheaper purchasing options, smuggling)
- Education and support for cessation
- Tobacco advertising and promotion

This report provides a detailed picture of the current tobacco control policy landscape in all six European countries, including cigarette smokers and e-cigarette users' beliefs, attitudes, and behaviours, following the passage of the TPD in 2014.

c. To compare smoking behaviour and the impact of policies between the 6 European **countries and other ITC countries.** The ITC Project aims to provide an evidence base to guide policies enacted under the FCTC, and to systematically evaluate the effectiveness of these legislative efforts. All ITC Surveys are developed using the same conceptual framework and methods, and the survey questions are designed to be identical or functionally equivalent in order to allow strong comparisons across countries. The evaluation studies conducted from the ITC Surveys take advantage of natural environments created when an ITC country implements a policy: changes in policy-relevant variables in that country from pre- to post-policy survey waves are compared to those in other ITC countries where that policy has not changed. This research design provides high levels of internal validity, allowing more confident judgments regarding the possible causal impact of the policy.

d. To suggest changes to current European tobacco policies. Recommendations to strengthen the current tobacco policies are made based on existing and derived survey information. The aim is to optimise the effects of tobacco control policies with regard to situational and individual difference moderators: (a) demographic variables; (b) personality variables (e.g. time perspective); (c) environmental context (e.g. number of peers/family members who smoke); and (d) the individual's smoking history (e.g. past quit attempts, smoking intensity and quitting smoking).

### **Survey Design** 1.3

The ITC 6E Survey is a longitudinal cohort study. In other words, the respondents who participate in this survey will be re-contacted in the future to participate in follow-up surveys. The respondents were recruited through a face-to-face multi-stage stratified random sample of the general population aged 18 or more.

### The Research Team

The ITC 6 European Country Survey is conducted by researchers throughout Europe from both the six participating countries as well as other institution partners within Europe and abroad.

| Investigators | Organization | Country |
|---|---|---|
| 1. Constantine Vardavas | European Network on Smoking and Tobacco Pre- | Belgium |
| (coordinator) | vention (ENSP) | |
| 2. Ann McNeill | Kings College London (KCL) | United Kingdom |
| 3. Ute Mons | German Cancer Research Center (DKFZ) | Germany |
| 4. Marc Willemsen | University of Maastricht (UniMaas) | Netherlands |
| 5. Yiannis Tountas | University of Athens (UoA) | Greece |
| 6. Antigona Trofor | Aer Pur Romania (APR) | Romania |
| 7. Brian Ward | European Respiratory Society (ERS) | Switzerland |
| 8. Geoffrey Fong | University of Waterloo (UW) | Canada |
| 9. Esteve Fernandez | Institut Català d'Oncologia (ICO) | Spain |
| 10. Tibor Demjén | Smoking or Health Hungarian Founation (SHFF) | Hungary |
| 11. Witold Zatonski | Health Promotion Foundation | Poland |
| 12. Aristidis Tsatsakis | University of Crete (UoC) | Greece |
| 13. Nicolas Bécuwe | Kantar Public Brussels (KP) | Belgium |

# 1.5 Country Timelines

Below are the timelines in conjunction with the tobacco control policies and ITC wave for each of the 6 countries.





Updated July 2016



# **GREECE**Timeline of Tobacco Control Policies and ITC Surveys

| .5 billion euros<br>Il price for most<br>30 per pack<br>pack | 2015 |
|---|---|
| cco products is 2<br>80% of total retai<br>bigarettes<br>cigarettes is €3.5<br>similar is €4 per | 2014 |
| 72014 Tax revenue for tobacco products is 2.5 billion euros Tax now represents 80% of total retail price for most optular pack of (20) eigarettes Lowest cost pack of oigarettes is €3.30 per pack Price of Mariboro or similar is €4 per pack | 2013 |
| N a | 2012 |
| July 2009 Comprehensive ban on smoking in enclosed spaces, workplaces, healthcare, food preparation, entertainment and other public and private areas. | 2011 |
| | 2010 |
| Dec 2008 Banned sale and advertising In health and educational acilities Banned sale of tobacco to minors (<18) Prohibited the manufacture of tems bearing resemblance to cobacco products | 2009 |
| Dec 2008 • Banned sale and advertising in intensity and educational facilities activities of the salidities of the salidities of the manufacture (items bearing resemblance to tobacco products | 2008 |
| <b>s</b><br>ification. | 2007 |
| Jan 2006 FCTC ratification. Isive | 2006 |
| July 2005 Comprehensive advertising ban enacted | 2005 |

Survey Mode: Personal (CAPI) Respondent Types: Smoker



23



# HUNGARY Timeline of Tobacco Control Policies and ITC Surveys

| 2014 Annual tax revenue from tobacco products is 1.3 million euros Annual tobacco control activity expenditure is £180,500 Tax represents 77% of total retail price of most popular cigarette brand pack Lowest cost pack of olgarettes (20) is £2.52 Price of Mariboro or similar is £3.46 |
|---|
| Sept 2012 • Enacted tobacco sale, licensing, and track & trace system. |
| Dec 2011 • Use of misleading terms banned • Enacted health warning legislation to comply with EU TPD (2001) |
| April 2004 • FCTC ratification Sept 2008 • All forms of promotion and sponsorship (direct/indirect) banned |
| Mandated tobacco products be sold in an area separated from unrelated products. Comprehensive smokefree legislation enacted - allowances made for select designated smoking areas smoking areas Smoking banned in private/public workplaces |
| Dec 1995 Comprehensive tobacco advertising ban 1999 Health warning legislation enacted: 30% front, 40% back, 10% sides and rotated warnings. Warnings must also appear at the point of sale Banned the sale of tobacco in social facilities and vending machines |

Updated July 2016



Survey Mode: Personal (CAPI) Respondent Types: Smoker



POLAND
Timeline of Tobacco Control Policies and ITC Surveys

| | 004 | <ul> <li>Health warnings</li> </ul> | mandated on smoked | tobacco products | <ul> <li>Required point of sale</li> </ul> | to display tobacco | | Sept Zuvo | | • Iviariulacture | product constin | alla ellissioni |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | March 2004 | <ul> <li>Health</li> </ul> | mandate | tobacco | <ul> <li>Require</li> </ul> | | health warnings | | 1 | \ | | |
| 200 | <ul> <li>Comprehensive</li> </ul> | advertising, promotion | and sponsorship ban | <ul> <li>Cessation helpline</li> </ul> | available | <ul> <li>Additives which increase</li> </ul> | risk of addiction banned | <ul> <li>Sale of tobacco to</li> </ul> | minors banned (<18) | <ul> <li>Prohibits self-serve</li> </ul> | tobacco sales (vending | machines) |

| 2014 | <ul> <li>Annual tax revenue is equal to 4.1 billion</li> </ul> | euros | <ul> <li>Government expenditure on tobacco</li> </ul> | control activity is equal to €225,000 | <ul> <li>Tax now represents 80.3% of total retail</li> </ul> | price for most popular pack of cigarettes | <ul> <li>Least expensive pack of oigarettes is €2.26</li> </ul> | <ul> <li>Pack of Marlboro or similar is €3.34</li> </ul> | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ealth warnings | ndated on smoked | acon products | equired point or sale | display tobacco | alth warnings<br>Sept 2006 | FCTC ratification | Manufacturers required to file list of all | product constituents, the reason for inclusion | and emission data - especially tar, nicotine | and CO for all brand variants |



Survey Mode: Personal (CAPI) Respondent Types: Smoker

Updated July 2016

54





# ROMANIA Timeline of Tobacco Control Policies and ITC Surveys

| 2016 • Excise tax placed on e-cigarette liquid starting at. 5 lei/mL (€.11) updated yearly to reflect inflation • Use of e-cigs prohibited wherever tobacco smoking is | 2016 |
|---|---|
| • Tax represents 75% of • Tax represents 75% of • total retail price for most popular peck of cigarettes • Lowest cost pack of cigarettes is equal to £2.85 • Pack of Marlboro or similar is equal to £3.32 • Government expenditure on tobacco control activity is equal to 4.5 million euros | 2014 |
| ill tobacco products: at teristics and position equired for olgarette mplemented ist of all product ist of all product is all brand variants anacted in all facilities a smoking areas on minors (-18) cks <20 units ducts via vending ucts banned | 2012 |
| Oct 2008 • Health warnings mandated on all tobacco products: at least 30% or packaging – characteristics and position specified • Pictorial and a combined 35% required for cigarette health warnings • Cigarette emission tolerances implemented • Manufacturers required to file list of all product constituents, the reason for inclusion and emission data – especially far, nicotine and CO for all brand wariants • Partial smoke-free legislation enacted in all facilities – allowances made for designated smoking areas • Banned the sale of cigarettes to minors (<18) • Banned the sale of cigarette packs <20 units • Banned the sale of tobacco products via vending machines • Marketing of oral tobacco products banned | 2010 |
| *Bupropion available with a prescription – cost covered by gov't *NT available in pharmacies without a prescription. Cost not covered by gov't *Smoking cessation programs available in some facilities where cost is fully covered *Jan 2008 *Comprehensive advertising, promotion and sponsorship ben | 2008 |
| 2007 • Vareniciine available with a prescription – cost covered by gov't • Smoking cessation helpline available Jan 2006 FCTC ratification | 2006 |
| 2004 • Minimum of 30 minutes broadcasted weekly for educational campaigns • Gov't ministries required to develop national education programs | 2004 |

Survey Mode: Personal (CAPI) Respondent Types: Smoker

09







Updated July 2016



# **SPAIN**Timeline of Tobacco Control Policies and ITC Surveys

| 2014 • Annual tax revenue for tobacco products is 7.1 billion euros • Tax represents 78% of total retail price for most popular pack of cigarettes popular pack of cigarettes is 2.95 • Pack of Mariboro or similar is £4.95 | 2014 |
|---|---|
| May 2010 Pictorial health warnings mandated | 2010 |
| Jan 2006 Discounted sale of tobacco prohibited Comprehensive smoke-free legislation enacted (Law 22/2008) – ellowances made for DSRs Sale of loose cigarettes and cigarillos or in packages <20 units prohibited Smoking or product placement in the media banned - Smoking or product placement in the media banned - Smoking an product placement in the dia banned - Match Group for the Prevention of Tobacco Addiction "established - Tobacco products and point of sale required to include reference to prohibition of sale to minors - Banned tobacco sale via vending machines, with exceptions | 2006 |
| Jan 2005<br>FCTC retification | 2005 |
| June 2003 • Comprehensive advertising promotion and sponsorship ban Sept 2003 • Prohibited the use of misleading descriptors Jan 2004 Olgarette emission tolerances implemented | 2004 |
| n all tobacco scrifted acrified d specific blined 35% for specified specific and repecific and repecific and repecific and repecific and repecified and repecified and repecified and repecified and repecified and repecified | 2003 |
| Oct 2002 - Health warnings mandated on all tobacco oppoudcts; at least 30% of primary surface—characteristics and position specified - Mandated rotating general and specific health warnings to cover a combined 38% for smoked tobacco products - 10% of cigarette package sides for emission data - Batch/lot numbers required - Sale of unpackage cigarettes prohibited - Manufacturers required to file list of all product constituents, the reason for inclusion and emission data — especially far, nicotine and CO for all brand variants | 2002 |



Survey Mode: Personal (CAPI) Respondent Types: Smoker and/or Dual User (Tobacco & E-Cig)



# Survey Process, Protocols and Fieldwork

### **Survey Process** 2.1

The ITC 6 European Country Wave 1 fieldwork was managed and coordinated by Kantar Public Brussels. The fieldwork was conducted in the 6 European countries by the following agencies: Foerster and Thelen (Germany), Metron Analysis (Greece), Kantar TNS Hoffman (Hungary), Kantar TNS Polska (Poland), Curs (Romania) and Kantar TNS Spain (Spain).

The ITC 6 European Country Wave 1 Survey fieldwork consisted of 7 main steps (see Appendix B). The interviewers:

- 1. Approached a household and introduced themselves;
- 2. Administered the Household Screener Survey to the Most Knowledgeable Individual (MKI);
- 3. Had each selected respondent read the information letter and obtained the respondent's consent:
- 4. Administered a survey screener to each selected respondent;
- 5. Completed the respondents' individual questionnaires;
- 6. Completed the individual outcome codes in the HRF/HEF Form B;
- 7. Thanked the respondents and provided a token of appreciation to the household. For each household of respondents, the respondent was presented with a token of appreciation of varying value dependent on the country as remuneration for their time (See Section 2.5 for remuneration amounts).

# Replenishment Participant Selection and Consent

**Identifying eligible members.** Adult cigarette smokers formed the only category of eligible respondents in a household.

**Selection of household members.** Household members aged 18 years and older were sampled. From households with cigarette smokers, up to one male and one female cigarette smoker were selected using the last birthday method of selection for each.

**Information and consent.** Once a respondent was selected, the information letter was provided and consent was administered to the respondent (See Appendix B).

### 2 SURVEY PROCESS, PROTOCOLS AND FIELDWORK

Table 1. Percentage of respondents who consented to take part in the second wave (Autumn 2017)

| Country | National Agency | Consenting<br>Respondents (%) |
|---------|---------------------------|-------------------------------|
| Germany | Foerster and Thelen | 93% |
| Greece | Metron Analysis | 69% |
| Hungary | Kantar TNS (TNS Hoffmann) | 60% |
| Poland | Kantar TNS (TNS Polska) | 70% |
| Romania | Curs | 95% |
| Spain | Kantar TNS Spain | 97% |

# 2.3 Household Screener Survey

In each selected household that contained eligible adult smokers, the identified key Informant or Most Knowledgeable Individual was given a brief Household Screener, from which respondents were selected. The purpose of the household screener was to identify residents of the household who fit the screening criteria of the project: (1)18 years or older; (2) smoke at least monthly.

If the Key Informant/Most Knowledgeable Individual was available at the first household visit, the Household Screener was administered, and then the individual household members were selected and interviewed if possible. If not, an appointment was made to come back to complete the Household Screener.

# 2.4 Main Questionnaire

### 2.4.1 Screeners

After completing the Household Screener and before administering the appropriate individual questionnaires, each selected respondent was given an individual survey screener. This screener confirms the information supplied by the Most Knowledgeable Individual at the individual level.

### 2.4.2 Content of Survey

A summary of the survey questions is given below:

- Demographic questions (e.g., age, gender, education, income, socio-economic status):
- Questions relevant to the policies of interest. These include measures of awareness (e.g., of warning labels, product ingredients, cessation assistance, advertising and promotion, prices, and e-cigarettes) and, where relevant, of more extensive cognitive processing (e.g., thinking about health warnings, relative harm between alternative products);
- Moderator variables (e.g., time perspective, stress, co-morbidities);
- Well-established questions assessing smoking behaviour;
- Other important psychosocial predictors of smoking behaviour (psychosocial mediating variables, e.g., normative beliefs, self-efficacy, intentions to quit).

### 2.4.3 Language of Survey

The survey questionnaire was translated into the national languages of all six participating countries: German; Greek; Hungarian; Polish; Romanian; and Spanish.

### 2.4.4 Length of the Interview

The survey was conducted by a face-to-face interview with the respondent. It took about 35 minutes to complete the survey questionnaire.

### 2.5 Remuneration

Interviewees were given the token of appreciation upon completion of the interview. Receipt of the token of appreciation was recorded by the interviewer as part of the post-interview section of the questionnaire. The interviewer had to confirm in the script that the respondent had received his or her voucher. Remuneration amounts in each country are listed in Table 2.

### 2 SURVEY PROCESS, PROTOCOLS AND FIELDWORK

Table 2. Remuneration amounts in each country

| Country | National Agency | Incentive (€) |
|---------|---------------------------|---------------|
| Germany | Foerster and Thelen | 10 |
| Greece | Metron Analysis | 5 |
| Hungary | Kantar TNS (TNS Hoffmann) | 10 |
| Poland | Kantar TNS (TNS Polska) | 10 |
| Romania | Curs | 7 |
| Spain | Kantar TNS Spain | 3 |

### 2.6 Progress Report

### 2.6.1 Survey Translation

All the surveys for Wave 1 fieldwork were finalized by the end of May 2016. Translation of the survey documents into the six national languages also took place over the course of the month of May. Translation was handled in house by the survey firm Kantar Public Brussels. The translation process used was the following: first the questionnaire was translated by an independent translator. Then this version was revised twice: first by an independent proof-reader and then by the national agency project manager. When the translation was finalised it was sent for approval to the national members of the Consortium who sent their final comments and agreements.

### 2.6.2 Field Work Preparation and Interviewer Training

The survey firm Kantar Public Brussels handled all fieldwork preparation within the six countries over the month of June 2016. Representatives from Kantar Public Brussels trained local country teams to use the tablet-based CAPI survey, as well as ensuring fieldwork operators followed the proper procedures outlined in the protocol.

### 2.6.3 Survey Fieldwork

The fieldwork started on June 16, 2016 and continued until September 12, 2016. Due to the international nature of the project, each country had varying start and completion dates. Table 3 outlines the fieldwork dates within each country.

| Country | National Agency | Fieldwork Dates |
|---------|---------------------------|----------------------|
| Germany | Foerster and Thelen | June 15–August 30 |
| Greece | Metron Analysis | June 16–September 12 |
| Hungary | Kantar TNS (TNS Hoffmann) | June 22–July 20 |
| Poland | Kantar TNS (TNS Polska) | June 25–August 11 |
| Romania | Curs | June 25–August 8 |
| Spain | Kantar TNS Spain | June 23–July 21 |

Table 3. ITC Europe fieldwork dates (2016).

Fieldwork in Athens, Greece had to be suspended for one week during the month of August (August 12 – August 19) due to much of the population being away in mid-August, a common vacation period. Fieldwork was concluded on September 12, 2016.

In Romania, extra call backs were conducted between September 2 and September 12 to ask BQ49221 (Q76.9) that could not be asked during the face-to-face survey. 789 respondents out of 1003 were reached and asked this question.

The total number of respondents completing the survey in each country and the size of the field work teams are listed in Tables 4 and 5, respectively.

| Table 4. Tota | l responden | ts completin | g the ITC Euro | pe Survey | in each country |
|---|---|---|---|---|---|

| Country | National Agency | # Completes |
|---------|---------------------------|-------------|
| Germany | Foerster and Thelen | 1003 |
| Greece | Metron Analysis | 1000 |
| Hungary | Kantar TNS (TNS Hoffmann) | 1000 |
| Poland | Kantar TNS (TNS Polska) | 1006 |
| Romania | Curs | 1001 |
| Spain | Kantar TNS Spain | 1001 |

### 2.6.4 Questionnaire Checking

The final version of the English questionnaire was checked by Kantar Public Brussels. Comments were sent to University of Waterloo and then the questionnaire was finalised. The master script of the questionnaire was then built. The script was checked by Kantar Public Brussels and sent for approval to the University of Waterloo.

Once the script was finalised in English, the national scripts were implemented and checked by national agencies before implementing the survey.

### 2 SURVEY PROCESS, PROTOCOLS AND FIELDWORK

| Country | National Agency | # Supervisors | # Interviewers |
|---------|---------------------------|---------------|----------------|
| Germany | Foerster and Thelen | 3 | 100 |
| Greece | Metron Analysis | 9 | 33 |
| Hungary | Kantar TNS (TNS Hoffmann) | 11 | 104 |
| Poland | Kantar TNS (TNS Polska) | 18 | 62 |
| Romania | Curs | 8 | 50 |
| Spain | Kantar TNS Spain | 4 | 24 |

Table 5. Size of the fieldwork team in each country

### 2.6.5 Data Checking and Cleaning

Once data checking was completed by Kantar Public Brussels, the data files were transferred securely to the University of Waterloo using an encrypted email and password sent by separate message.

Once the data were successfully transferred, the University of Waterloo data analyst commenced data cleaning. The data analyst conducted duplicate entry comparisons of the data files, using the SAS statistical software and identified discrepancies between the two data files. A list of these discrepancies were sent to the Kantar Public Brussels data manager for verification and correction. The Kantar Public Brussels data manager sent the corrections to the University of Waterloo data analyst for verification.

After discrepancies had been identified and corrections sent by the Kantar Public Brussels data manager, the University of Waterloo data analyst conducted additional checks on the data to ensure that all skip patterns had been correctly followed and to ensure that the data did not contain invalid values. Respondent identifier codes were also checked thoroughly to ensure the data could be correctly linked within a survey wave and between waves over time. Any additional discrepancies that were identified were also sent back to the in-country data manager for verification. This back and forth communication between the University of Waterloo data analyst and the Kantar public Brussels data manager went on until the data were deemed clean by the University of Waterloo data analyst. Following data processing and cleaning, sampling weights were constructed for the dataset and the final, cleaned datasets were released to the country team, by posting them on the secure, internal ITC website.

### 2.6.6 Data Delivery

Wave 1 data were delivered to the Data Management Centre (DMC) at the University of Waterloo on October 4, 2016. A DMC data analyst processed the Wave 1 data which were released in January 2017 and have been available for further analysis.

### **Monitoring and Quality Control** 3

### **Management of Fieldwork Teams** 3.1

The project fieldwork team consisted of five levels of management, including:

- **Project Manager:** responsible for overseeing all aspects of the survey fieldwork (design of the survey, sampling design and central briefing of national project managers), as well as administrative duties and communicating with the ITC Six European Country team in Waterloo and the Project Consultants.
- Fieldwork Manager: responsible for managing the survey fieldwork in all 6 countries, setting up the central coordination of fieldwork (supply sample, load script), ensuring the daily communication with national project manager and applying quality control on a regular basis.
- Project Manager (Fieldwork): responsible for managing national fieldwork including checking national script, data quality control and proving weekly reporting on fieldwork progress.
- Field Supervisors: responsible for supervising the interviewers, contacting local authorities and monitoring the interviews.
- Interviewers: responsible for obtaining consent, interviewing respondents, and reporting to the field supervisor with any problems.

### 3.2 **Survey Protocol**

An English survey protocol outlining the process in which fieldwork was to be conducted was written to ensure a benchmark standard for fieldwork across each country. The survey firm, Kantar Public Brussels, relayed the information outlined in the survey protocol to the country teams developing a survey wave manual that was used for a central briefing

### **Monitoring and Quality Assurance** 3.3

To ensure the accuracy and quality of the ITC Six European Country Survey, the survey fieldwork was monitored in several ways.

• Centralised data management: The fieldwork was centrally managed by Kantar Public Brussels. Data were centrally transmitted via NFIELD software and therefore Kantar Public Brussels were able to assess progress and access data on a regular basis.

### 3 MONITORING AND QUALITY CONTROL

- **Progress Reports:** The Project Manager was provided regular progress reports on completion rates and any problems or issues by the survey firm, Kantar Public Brussels. Those reports were then presented to the Data Management team on a weekly basis.
- **Field Supervision:** The Field Supervisor was in charge of supervising the interviewers, helping them when they had a question regarding the contact procedure, the methodology or the script and liaising with the national agency.
- **Identification Numbers:** Identification numbers would be generated automatically by the CAPI program. All interviews in the six countries were conducted on Tablets using the NFIELD software.
- Quality control at local level: 10% back checks on interviews conducted within a week of completion (national institutes). Checks on coding (at least 10% of answers recoded as part of overall quality back check). Comparison between raw samples and national universe (central team). Ensuring item response is 100% within each completed survey

## 3.4 Handling Special Situations

**Private interviews.** Adult participants were interviewed alone whenever possible. If another person insisted on being present, the respondent needed to agree for the interview to proceed.

**Proxy interviews.** A proxy interview is an interview conducted with another knowledgeable member of the household on behalf of the selected respondent. Proxy interviews were *not allowed* in the ITC Six European Country Survey.

**Respondent not available.** If a respondent was unavailable, an appointment time (hard appointment) was rescheduled to interview that respondent.

**Substitution.** Only if a selected household was recorded to have the disposition "No one at home" or "Cannot answer" for all four visits over four different times, (weekday day-time, weekday nighttime, weekend day-time and weekend night-time) could the household be replaced by a substitute, selected by the Field Supervisor.

**Handling multiple respondents.** An interviewer could not interview two adults at the same time.

# Sampling Design and Weight Construction

### Sampling design 4.1

The ITC 6E Survey is a prospective longitudinal study, and its sampling design was chosen to yield nationally representative random samples of adult smokers residing in Germany, Greece, Hungary, Poland, Romania and Spain. Respondents were interviewed between June 18 and September 12, 2016. All interviews were conducted face-to-face by interviewers using tablets (CAPI).

To qualify for the study, respondents had to be 18 years old or more, smoke at least monthly, and have smoked more than 100 cigarettes in their lives. In each country, a probability sample of dwellings was approached. At each dwelling, an informant was identified and asked the number of male smokers of at least 18 years of age and the number of female smokers of at least 18 years of age. Where possible a male smoker and a female smoker were selected from each household, using the Next Birthday method (Binson & Catania (2000)). No substitution within a household was allowed, except when it was known that the selected respondent would be absent for the entire fieldwork period.

The probability sample of dwellings was chosen as follows in each country. The country was divided into major geographic regions, namely NUTS2 regions for all countries except Germany, where NUTS1 regions were used. (Excluded for Greece were the islands in the Ionian Sea, the northern Aegean Sea and the southern Aegean Sea; excluded for Spain were the Canaries, Ceuta and Melilla.) The geographic strata were the NUTS regions crossed with degree of urbanization (urban, intermediate, rural). The strata were conceptually considered to be a union of clusters, each the size of an enumeration area, with the objective of sampling 100 clusters per country, and obtaining 10 adult smokers in each cluster. Clusters were allocated to strata proportionally to 18+ population size, subject to requiring at least two clusters in each stratum, and selected at random within each stratum.

In each selected cluster, a random walk method was to be used to select dwellings. A starting point was to be chosen at random using GPS coordinates, and a random walk path predrawn on a tablet; the interviewers were to follow the path and approach every fifth address on the path, for household screening and potential selection of adult smokers for interview. If an address corresponded to multiple households, a single household was to be selected at random. For each chosen address, contact was attempted up to four times.

As indicated above, one randomly selected male smoker and one randomly selected female smoker were to be selected for interview from a household where possible. Screening of households was to continue until the required number of smokers from the cluster had been interviewed.

The ITC 6E Wave 1 sample has the following sample sizes. Appendix A provides a detailed breakdown of the sample size within each country by sampling region, degree of urbanization and sex-age group.

### 4 SAMPLING DESIGN AND WEIGHT CONSTRUCTION

Table 6. Country sample sizes

| Country | Sample Size |
|---------|-------------|
| Germany | 1003 |
| Greece | 1000 |
| Hungary | 1000 |
| Poland | 1006 |
| Romania | 1001 |
| Spain | 1001 |
| Overall | 6011 |

## 4.2 Weight construction

### 4.2.1 General comments about weight construction

As with most survey weights, the ITC 6E Wave 1 weights are constructed to correct and adjust for sample misrepresentation caused by unequal sampling probabilities, frame error (i.e., under-coverage and multiplicity), and non-response, as well as to improve precision of estimates through the use of auxiliary information (e.g., smoking prevalences). We briefly describe these key concepts of weight construction in this section, but refer the reader to Levy & Lemeshow (2008), chapter 16, for more detailed information.

Basic design weights are defined as the reciprocals of selection probabilities, and thus adjust for sample misrepresentation caused by unequal sampling probabilities. For example, a smoker residing alone has a probability of selection twice that of a smoker residing with another smoker of the same sex, and thus will typically have a smaller weight to compensate.

The sampling frame is effectively a set of starting points within selected areas of each stratum, and may fail to cover some addresses. This is referred to as frame under-coverage, and can result in non-coverage bias. To reduce non-coverage bias in the ITC 6E Survey, post-stratification adjustments have been performed on the sampling weights to ensure that, for each stratum/sex/age group, the totals of the sampling weights are approximately equal to assumed benchmarks; see step 3 in section 4.2.2. Note that these benchmark figures are also referred to as calibration or target figures, and thus the post-stratification adjustment is also referred to as weight calibration.

If non-respondents behave differently than respondents, then inference based solely on the sample of respondents will be biased unless adjustments are made. The greater the expected proportion of non-response, the greater this bias is likely to be. In the ITC 6E Survey, the post-stratification adjustments described in the above paragraph also adjust for non-response bias. It should be noted that if data are missing completely at random (MCAR, see

Little & Rubin (2002)) within each stratum/sex/age group, then non-response bias will be completely eliminated. Realistically, however, non-response bias is reduced but not eliminated by calibration in the ITC 6E Survey.

It is well known, from survey sampling theory, that in the vast majority of cases, the ratio estimator of a population total has much greater precision than the commonly used Horvitz-Thompson estimator. Heuristically, this is due to the fact that the ratio estimator utilizes auxiliary (i.e., additional) information in addition to the sampling weights, whereas the Horvitz-Thompson estimator does not. As mentioned above, benchmark figures have been used to calibrate the ITC 6E sampling weights in order to reduce biases from frame errors and non-response. A consequence of using this auxiliary information in weight computation is that the precision of most estimates is increased. The calibrating procedure yields so-called ratio weights, which enable all estimators to inherit the increased precision of the ratio estimator.

### 4.2.2 Wave 1 weights

Within each country, computation of sampling weights for the smokers who completed the Wave 1 survey proceeded as follows.

Step 1: Each respondent i was assigned an initial weight  $w_i^{(1)}$ , which can be viewed as an adjustment for the probability of selection within a given household. Formally, the  $w^{(1)}$  weights are given by

$$w_i^{(1)} = \frac{\text{\#18+ smokers of same sex as } i \text{ in household}}{\text{\#18+ smokers interviewed of same sex as } i \text{ in household}}$$

Note that the denominator should be 1 by design; as well, #18+ smokers of same sex as i in household was capped at 4 to prevent large households from having undue influence on the weights.

Step 2: Traditionally in two stage designs, the primary sampling units (psus) correspond to fixed geographic areas, and are sampled with probability proportional to size. Then approximately the same number of dwelling addresses is chosen at random in each psu, giving approximately equal inclusion probabilities for households. Traditionally we compute the household inclusion probability within a stratum and psu more precisely, and take the reciprocal as the household weight, but it is not a very bad approximation to take all sample households within a stratum to have the same "raising factor", and the inclusion probabilities of individuals within strata to be approximately proportional to their inclusion probabilities within households.

In the case of the random walk design, the probability of inclusion of a dwelling or household is the proportional to the number of random walks in which it would

### 4 SAMPLING DESIGN AND WEIGHT CONSTRUCTION

be one of the sampled households. It cannot be computed from the information available, and thus we have taken the inclusion probabilities of households to be approximately equal within strata, and the inclusion probabilities of individuals within strata to be approximately proportional to their inclusion probabilities within households.

Step 3: A post-stratification adjustment was then performed to calibrate the  $w_i^{(1)}$  weights to smoking prevalence by stratum/sex/age groups. We used the same categories as used in the Eurobarometer surveys. To this end, age was divided into 3 intervals (i.e., [18, 39), [40, 54), and 55+); urbanization was divided into 3 categories: rural (U1), intermediate (U2), and cities/large urban area (U3).

Eurobarometer survey data from 2014 were used to model smoking prevalence, using a weighted logistic regression of smoking status (binary) on sex, age group, urbanization and NUTS region. A sex  $\times$  age group interaction was also included. This yielded an estimated probability of being a smoker

for someone with sex s, age group a, urbanization u and region r. (For this purpose, in Spain, Navarra and Basque Country were put together, as were Rioja and Aragon; in Germany, Bremen and Niedersachsen were put together; in each case, it was because the smaller region had no smoker respondents in the Eurobarometer survey. In Spain, the smoking rate for Cantabria, with no Eurobarometer respondents, was taken to be the average of the rates for Galicia and Asturias.)

The logistic regression analysis was restricted to Eurobarometer respondents aged 18 and older.

Projections from census data for January 1, 2015, found at the Eurostat website (see the tables in Appendix B), were used to estimate

$$N(s, a, u, r)$$
,

the number of people of sex s, age group a, urbanization u and region r. Specifically, there are tables for:

- (a) Population for each region (NUTS2), age (18+, by single year age category) and sex
- (b) Number of households by region (NUTS2) by degree of urbanization

For Germany, it was possible to obtain the figures for the NUTS1 regions instead.

Using (b), and making the assumption that the population of individuals follows the distribution of households by urban/intermediate/rural areas, it was possible to multiply total population estimates for (a) by the proportion of the population in

each urban category to obtain population estimates within the 4-way table needed for calibration (region  $\times$  urbanization  $\times$  sex  $\times$  age).

The degree of urbanization is not available on the Eurobarometer data for Germany; a different classification is used, as follows, where "Kern" = core and "Rand" = edge.

- Kern  $\geq$  500,000
- Rand  $\geq 500,000$
- Kern 100,000–500,000
- Rand 100,000–500,000
- Kern 50,000–100,000
- Rand 50,000–100,000
- 20,000-50,000
- 5000-20,000
- 2000-5000
- < 2000

Eurostat defines urban areas as areas where the majority of the population lives in an urban centre of at least 50,000 people. Thus, in the Eurobarometer data, when carrying out the logistic regression for Germany, the Kern areas were classified as urban, the Rand areas as intermediate, and the rest as rural.

To estimate the number of smokers S(s, a, u, r) in a cell defined by sex crossed with age group, crossed with urbanization crossed with region, N(s, a, u, r) was multiplied by p(s, a, u, r).

See Appendix B for the tables of the estimated population sizes N(s, a, u, r), and the estimated numbers of smokers in each S(s, a, u, r).

Some cells C(s, a, u, r) were merged so that the number of ITC respondents in each cell would be not too small; see Appendix A. Accordingly, let the final set of merged cells for a country be denoted by C(k), k = 1, ..., K, and let the estimated number of smokers in the population in cell C(k) be denoted by S(k), which is the sum of S(s, a, u, r) over all of the original cells C(s, a, u, r) in the merged cell C(k).

For respondents in cell C(k), the post-stratification adjustment consisted in multiplying their  $w_i^{(1)}$  weights by a factor to produce calibrated  $w_i^{(2)}$  "inflation weights". The inflation weight for respondent i is interpreted as the number of people in the population represented by that respondent. These inflation weights are such that their sum over all respondents in a cell C(k) is equal to the estimated number of adult smokers in that cell. Formally, if i is in cell C(k),

$$w_i^{(2)} = w_i^{(1)} \times \frac{S(k)}{\sum_{i \in c(k)} w_i^{(1)}},$$

where c(k) is the set of all respondents in cell C(k). The inflation weights are variable "aDE49915v" in the data set.

### 4 SAMPLING DESIGN AND WEIGHT CONSTRUCTION

Step 4: To facilitate comparisons among the 6 countries and with other ITC countries, the  $w_i^{(2)}$  weights were rescaled to have a mean equal to 1 in each country. This yielded the "analytic"  $w_i^{(3)}$  weights, which are formally defined as

$$w_i^{(3)} = w_i^{(2)} \times \frac{n_{\gamma}}{\sum_{i \in S_{\gamma}} w_i^{(2)}},$$

where  $S_{\gamma}$  is the set of all sampled smokers in country  $\gamma$ , and  $n_{\gamma}$  is the size of that sample from Table 1.

Hence, in each country  $\gamma$ , the  $w_i^{(3)}$  weights sum to  $n_\gamma$ . The analytic weights are variable "aDE49919v" in the data set.

The means and coefficients of variation (CVs) of the inflation weights in the six countries are given in Appendix C.

### 4.3 Taking the sampling design into account in analyses

The inflation weights and analytic weights adjust for sampling bias in the estimation of population means, ratios, regression coefficients, and more generally parameters that are defined as the solutions of population level estimating equations. Analyses of the data should also take into account the fact that the sampling design within each country is both stratified (tending to increase efficiency) and two-stage at the household level (tending to decrease efficiency because the sample is clustered in primary sampling units (PSUs). The statistical software packages SAS, SPSS, Stata, R and SUDAAN are able to produce standard errors and hypothesis tests for basic analyses that account for the complex sampling design. In each case, the software requires the stratum and PSU variables and the weight variable to be specified.

### 4.3.1 Specification of strata and PSUs for analyses

In the ITC 6E sampling design, in each of the countries there was at least one stratum with a single or "lonely PSU". In such a case, there is no design-based unbiased estimator of the variance of a linear estimator, such as an estimator of a population mean. Some software packages, such as SAS, will simply omit from the analysis data from a stratum with a single PSU. This makes the analysis representative only of the remaining strata. Other packages, such as SUDAAN, use a model-based assumption to allow the single-PSU stratum to contribute to the overall estimation of variance.

An alternative way of handling this situation is to collapse strata, most simply to merge each single-PSU stratum with another that is geographically close to it and can be expected to
have similar attributes. This choice of strata to merge is motivated by the need not to lose too much of the advantage of stratification: if the two strata being merged have very different means, for example, the merging will make the standard error estimation blind to the efficiency gain from the original stratification, meaning that standard errors will tend to be overestimated.

With the ITC 6E data, we have used the stratum collapsing technique, where possible merging a single-PSU stratum with another which is within the same NUTS region and has the same level of urbanization. The variable name for the collapsed strata or "variance strata" is "VARSTRAT". The variable name for PSU is "VARPSU".

### 4.3.2 Bootstrap weights

In another approach to accounting for the complex sampling design, we have provided a set of bootstrap weights, based on the Rao and Wu (1988) bootstrap technique, and constructed as follows.

For b = 1, ..., 6000, we produced a b-th "column" of initial bootstrap weights, as follows. Within each variance stratum h as defined in Section 3.1, if there are  $n_h$  sampled PSUs, we selected  $n_h$  PSUs by simple random sampling with replacement. For each respondent (h, i, j) in sampled PSU (h, i), that person's bootstrap weight  $w_{hijb}$  is the main (inflation or analytic) weight  $w_{hij}$  times  $[1 - \lambda_{1h} + (\text{number of times PSU } (h, i) \text{ has been "resampled"}) \times$  $\lambda_{1h}$ ], where  $\lambda_{1h} = \sqrt{n_h/n_h-1}$ . The bootstrap weight  $w_{hijb}$  will be 0 if (h,i) was not resampled, 1 if (h, i) was resampled once, a higher number if (h, i) was resampled twice, and so on.

The columns of initial bootstrap weights were then averaged, 12 at a time, to produce 500 averaged bootstrap weight variables. In the data set, the averaged analytic bootstrap weights are named "RSBSW001" to "RSBSW500".

Because of the fine stratification of the survey design, calibration of each of the initial 6000 bootstrap weight columns with the same method as for the main weights was not feasible. At the same time, it was found that calibration of the averaged bootstrap weights led to underestimation of standard errors as compared with the output of linearization methods. Thus neither the original 6000, nor the 500 averaged bootstrap weights which are provided with the data, have been calibrated.

The averaged bootstrap weights can be used with complex survey software to produce standard errors for various parameter estimates. Typically a BRR (balanced repeated replication) option is used, because the formula for producing standard errors with BRR is easily translated into the formula for producing standard errors in bootstrapping. A useful document is "Weighted estimation and bootstrap variance estimation for analyzing survey data: How to implement in selected software", by Gagné, Roberts and Keown, at http:

#### REFERENCES

//www.statcan.gc.ca/pub/12-002-x/2014001/article/11901-eng.htm. The paper by Phillips (2004) explaining the Fay adjustment is available at http://www5.statcan.gc.ca/olc-cel/olc. action?ObjId=12-002-X20040027032&ObjType=47&lang=en&limit=0.

## References

- Binson, D. & Catania, J. A. (2000), Random selection in a national telephone survey: a comparison of the Kish, next-birthday and last-birthday methods. Journal of Official Statistics, 16, 53-60.
- Levy, P. S. & Lemeshow, S. (2008), Sampling of Populations: Methods and Applications, 4 edn, John Wiley & Sons, Hoboken, NJ.
- Little, R. J. A. & Rubin, D. B. (2002), Statistical Analysis with Missing Data, 2 edn, John Wiley & Sons, Hoboken, NJ.
- Phillips, O. (2004), Using bootstrap weights with WesVar and SUDAAN. Research Data Centres, Information and Technical Bulletin, 1(2), 6-15.
- Rao, J. N. K. & Wu, C. F. J. (1988), Resampling inference with complex survey data. *Journal of* the American Statistical Association, 83, 231-241.

## **Appendices**

## Sample size tables

A detailed set of sample size tables are available upon request that depict the total number of respondents sampled in each country. Sample sizes in these tables are broken down by sampling region crossed with degree of urbanization crossed with sex and age group.

#### Benchmark/calibration figures B

The following tables show (a) the population estimates as of 2015-01-01 and (b) the estimated numbers of smokers in each country for region crossed with urbanization crossed with sex and age group.

Projections from census data for January 1, 2015, found at the Eurostat website were used to estimate the population numbers the number of people by region, urbanization, sex and age group. Specifically, there are tables for:

- (a) Population for each region (NUTS2), age (18+, by single year age category) and sex http://ec.europa.eu/eurostat/web/population-demography-migration-projections/ population-data/database
- (b) Number of households by region (NUTS2) by degree of urbanization http://ec.europa.eu/eurostat/web/degree-of-urbanisation/data/database
  - the number of households table can be found under the "Labour market" category.

Using (b), and making the assumption that the population of individuals follows the distribution of households by urban/intermediate/rural areas, it was possible to multiply total population estimates for (a) by the proportion of the population in each urban category to obtain population estimates within the 4-way table needed for calibration (region × urbanization  $\times$  sex  $\times$  age).

## Germany

Table 7. Total population by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| Schleswig-Holstein | 89,810 | 87,488 | 121,525 | 88,173 | 88,563 | 142,914 |
| Hamburg | 274,315 | 202,824 | 235,560 | 282,872 | 196,011 | 289,967 |
| Niedersachsen | 265,469 | 244,947 | 333,752 | 253,669 | 243,232 | 392,266 |
| Bremen | 97,618 | 73,888 | 100,530 | 92,860 | 70,766 | 124,587 |
| Nordrhein-Westfalen | 1,177,584 | 1,041,964 | 1,375,304 | 1,150,138 | 1,037,419 | 1,662,517 |
| Hessen | 270,246 | 237,373 | 308,814 | 264,987 | 233,977 | 362,859 |
| Rheinland-Pfalz | 115,782 | 104,617 | 145,384 | 111,442 | 104,290 | 169,752 |
| Baden-Württemberg | 417,631 | 349,509 | 450,890 | 398,497 | 343,131 | 531,690 |
| Bayern | 537,151 | 458,523 | 586,202 | 517,025 | 449,289 | 691,057 |
| Saarland | 25,204 | 22,735 | 34,895 | 23,762 | 23,029 | 41,664 |
| Berlin | 542,185 | 391,150 | 486,701 | 542,693 | 373,367 | 594,783 |
| Brandenburg | 48,060 | 51,624 | 76,003 | 44,112 | 50,030 | 89,600 |
| Mecklenburg-Vorpommern | 68,580 | 63,800 | 98,515 | 61,356 | 60,730 | 118,671 |
| Sachsen | 214,326 | 182,593 | 296,109 | 192,249 | 170,417 | 369,170 |
| Sachsen-Anhalt | 73,862 | 71,255 | 112,825 | 64,832 | 67,739 | 139,879 |
| Thüringen | 64,046 | 59,214 | 93,642 | 56,682 | 55,864 | 113,583 |
| Intermediate | | | | | | |
| Schleswig-Holstein | 165,733 | 161,447 | 224,258 | 162,711 | 163,431 | 263,728 |
| Hamburg | 0 | 0 | 0 | 0 | 0 | 0 |
| Niedersachsen | 413,021 | 381,092 | 519,257 | 394,663 | 378,424 | 610,294 |
| Bremen | 0 | 0 | 0 | 0 | 0 | 0 |
| Nordrhein-Westfalen | 953,646 | 843,816 | 1,113,766 | 931,419 | 840,136 | 1,346,360 |
| Hessen | 409,976 | 360,106 | 468,485 | 401,998 | 354,955 | 550,474 |
| Rheinland-Pfalz | 239,400 | 216,313 | 300,606 | 230,426 | 215,637 | 350,992 |
| Baden-Württemberg | 799,584 | 669,159 | 863,260 | 762,950 | 656,948 | 1,017,957 |
| Bayern | 708,877 | 605,112 | 773,609 | 682,316 | 592,926 | 911,986 |
| Saarland | 80,055 | 72,214 | 110,838 | 75,474 | 73,147 | 132,336 |
| Berlin | 0 | 0 | 0 | 0 | 0 | 0 |
| Brandenburg | 133,172 | 143,047 | 210,603 | 122,233 | 138,631 | 248,278 |
| Mecklenburg-Vorpommern | 47,367 | 44,066 | 68,044 | 42,378 | 41,946 | 81,965 |
| Sachsen | 203,110 | 173,037 | 280,613 | 182,188 | 161,498 | 349,850 |
| Sachsen-Anhalt | 92,217 | 88,962 | 140,863 | 80,943 | 84,573 | 174,641 |
| Thüringen | 105,514 | 97,552 | 154,272 | 93,381 | 92,033 | 187,123 |
| Rural | | | | | | |
| Schleswig-Holstein | 88,178 | 85,898 | 119,316 | 86,570 | 86,953 | 140,316 |
| Hamburg | 0 | 0 | 0 | 0 | 0 | 0 |
| Niedersachsen | 319,397 | 294,707 | 401,552 | 305,201 | 292,643 | 471,953 |
| Bremen | 0 | 0 | 0 | 0 | 0 | 0 |
| Nordrhein-Westfalen | 197,041 | 174,348 | 230,125 | 192,449 | 173,588 | 278,183 |
| Hessen | 139,175 | 122,246 | 159,037 | 136,466 | 120,497 | 186,870 |
| Rheinland-Pfalz | 163,695 | 147,909 | 205,546 | 157,559 | 147,447 | 239,998 |
| Baden-Württemberg | 273,799 | 229,138 | 295,603 | 261,255 | 224,957 | 348,576 |
| Bayern | 512,235 | 437,254 | 559,010 | 493,042 | 428,449 | 659,002 |

Table 7. (Continued)

| | | Men | | Women | | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Saarland | 19,433 | 17,529 | 26,905 | 18,321 | 17,756 | 32,124 |
| Berlin | 0 | 0 | 0 | 0 | 0 | 0 |
| Brandenburg | 99,019 | 106,361 | 156,591 | 90,885 | 103,078 | 184,604 |
| Mecklenburg-Vorpommern | 83,169 | 77,373 | 119,473 | 74,409 | 73,649 | 143,916 |
| Sachsen | 103,424 | 88,111 | 142,889 | 92,771 | 82,236 | 178,145 |
| Sachsen-Anhalt | 102,924 | 99,292 | 157,218 | 90,342 | 94,393 | 194,918 |
| Thüringen | 97,939 | 90,549 | 143,197 | 86,677 | 85,426 | 173,689 |

Table 8. Total smokers by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| Schleswig-Holstein | 70,941 | 74,898 | 84,788 | 60,637 | 63,172 | 76,245 |
| Hamburg | 104,925 | 100,378 | 64,873 | 75,301 | 56,980 | 45,960 |
| Niedersachsen | 72,924 | 91,782 | 62,946 | 46,041 | 48,744 | 40,521 |
| Bremen | 26,816 | 27,686 | 18,960 | 16,854 | 14,182 | 12,870 |
| Nordrhein-Westfalen | 469,974 | 533,902 | 398,288 | 322,154 | 316,828 | 279,469 |
| Hessen | 96,235 | 110,758 | 78,253 | 64,816 | 62,682 | 52,252 |
| Rheinland-Pfalz | 43,268 | 50,802 | 38,963 | 28,852 | 29,524 | 26,074 |
| Baden-Württemberg | 127,586 | 143,404 | 95,859 | 81,652 | 77,376 | 62,739 |
| Bayern | 187,681 | 210,645 | 145,319 | 123,724 | 117,804 | 97,024 |
| Saarland | 11,370 | 12,852 | 11,700 | 7,723 | 8,113 | 8,333 |
| Berlin | 239,863 | 217,714 | 159,346 | 172,142 | 128,550 | 115,626 |
| Brandenburg | 14,951 | 21,512 | 13,985 | 9,224 | 11,512 | 10,815 |
| Mecklenburg-Vorpommern | 32,651 | 37,629 | 35,268 | 21,315 | 22,804 | 25,692 |
| Sachsen | 60,333 | 69,860 | 57,386 | 35,874 | 35,089 | 39,317 |
| Sachsen-Anhalt | 38,076 | 44,698 | 44,566 | 24,889 | 27,990 | 34,186 |
| Thüringen | 26,893 | 31,608 | 28,795 | 16,874 | 18,094 | 20,490 |
| Intermediate | | | | | | |
| Schleswig-Holstein | 124,913 | 133,807 | 146,328 | 104,444 | 109,417 | 127,117 |
| Hamburg | 0 | 0 | 0 | 0 | 0 | 0 |
| Niedersachsen | 97,308 | 124,922 | 82,614 | 60,344 | 64,105 | 52,302 |
| Bremen | 0 | 0 | 0 | 0 | 0 | 0 |
| Nordrhein-Westfalen | 334,634 | 388,999 | 277,439 | 224,006 | 221,376 | 190,106 |
| Hessen | 127,257 | 149,768 | 101,380 | 83,857 | 81,462 | 66,277 |
| Rheinland-Pfalz | 78,236 | 93,988 | 69,019 | 51,016 | 52,443 | 45,173 |
| Baden-Württemberg | 210,770 | 241,968 | 155,473 | 132,219 | 125,806 | 99,963 |
| Bayern | 215,640 | 247,430 | 163,618 | 139,056 | 133,053 | 106,976 |
| Saarland | 32,086 | 37,132 | 32,265 | 21,246 | 22,449 | 22,378 |
| Berlin | 0 | 0 | 0 | 0 | 0 | 0 |
| Brandenburg | 35,783 | 52,598 | 38,751 | 21,647 | 27,116 | 24,952 |
| Mecklenburg-Vorpommern | 20,136 | 23,760 | 21,243 | 12,807 | 13,783 | 15,049 |
| Sachsen | 49,112 | 58,019 | 45,936 | 28,676 | 28,133 | 30,927 |
| Sachsen-Anhalt | 42,789 | 51,420 | 48,879 | 27,237 | 30,810 | 36,395 |
| Thüringen | 39,209 | 47,059 | 40,959 | 23,952 | 25,815 | 28,424 |
| Rural | , | ., | -, | -, | -,- | -, |
| Schleswig-Holstein | 66,521 | 71,244 | 77,973 | 55,647 | 58,285 | 67,773 |
| Hamburg | 0 | 0 | 0 | 0 | 0 | 0 |
| Niedersachsen | 75,474 | 96,870 | 64,088 | 46,818 | 49,749 | 40,588 |
| Bremen | 0 | 0 | 0 | 0 | 0 | 0 |
| Nordrhein-Westfalen | 69,319 | 80,549 | 57,508 | 46,419 | 45,879 | 39,419 |
| Hessen | 43,311 | 50,964 | 34,527 | 28,562 | 27,738 | 22,574 |
| Rheinland-Pfalz | 53,643 | 64,400 | 47,337 | 34,994 | 35,962 | 30,984 |
| Baden-Württemberg | 72,392 | 83,063 | 53,415 | 45,432 | 43,214 | 34,335 |
| Bayern | 156,232 | 179,187 | 118,622 | 100,827 | 96,444 | 77,630 |

Table 8. (Continued)

| | | Men | | Women | | |
|------------------------|--------|--------|--------|--------|--------|--------|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Saarland | 7,808 | 9,031 | 7,854 | 5,172 | 5,464 | 5,448 |
| Berlin | 0 | 0 | 0 | 0 | 0 | 0 |
| Brandenburg | 26,686 | 39,205 | 28,907 | 16,150 | 20,224 | 18,627 |
| Mecklenburg-Vorpommern | 35,438 | 41,797 | 37,395 | 22,553 | 24,267 | 26,509 |
| Sachsen | 25,080 | 29,623 | 23,462 | 14,649 | 14,375 | 15,801 |
| Sachsen-Anhalt | 47,860 | 57,490 | 54,696 | 30,481 | 34,472 | 40,757 |
| Thüringen | 36,394 | 43,771 | 38,133 | 22,302 | 24,030 | 26,470 |

## Greece

Table 9. Total population by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| Attica | 388,620 | 294,972 | 383,376 | 391,428 | 332,028 | 492,459 |
| Crete | 35,095 | 25,632 | 33,455 | 35,762 | 25,951 | 38,171 |
| Eastern Macedonia & Thrace | 8,468 | 5,743 | 9,028 | 7,477 | 6,016 | 10,782 |
| Central Macedonia | 100,134 | 80,723 | 114,028 | 102,259 | 85,395 | 138,160 |
| Western Macedonia | 0 | 0 | 0 | 0 | 0 | 0 |
| Epirus | 9,536 | 7,980 | 14,266 | 10,123 | 7,910 | 15,892 |
| Thessaly | 43,794 | 35,618 | 57,173 | 43,497 | 36,106 | 65,792 |
| Western Greece | 31,676 | 23,520 | 34,974 | 30,516 | 23,489 | 39,965 |
| Central Greece | 6,870 | 5,568 | 8,244 | 6,143 | 5,255 | 9,420 |
| Peloponnese | 9,437 | 7,952 | 13,010 | 8,738 | 7,937 | 14,038 |
| Intermediate | | | | | | |
| Attica | 138,647 | 105,236 | 136,776 | 139,649 | 118,457 | 175,693 |
| Crete | 17,383 | 12,696 | 16,571 | 17,714 | 12,854 | 18,907 |
| Eastern Macedonia & Thrace | 41,523 | 28,160 | 44,269 | 36,663 | 29,497 | 52,867 |
| Central Macedonia | 86,363 | 69,622 | 98,347 | 88,196 | 73,651 | 119,160 |
| Western Macedonia | 17,623 | 15,868 | 24,119 | 17,586 | 15,843 | 26,518 |
| Epirus | 8,626 | 7,219 | 12,906 | 9,157 | 7,156 | 14,376 |
| Thessaly | 21,626 | 17,589 | 28,233 | 21,479 | 17,830 | 32,489 |
| Western Greece | 23,500 | 17,450 | 25,947 | 22,640 | 17,426 | 29,650 |
| Central Greece | 28,319 | 22,954 | 33,985 | 25,324 | 21,664 | 38,832 |
| Peloponnese | 23,304 | 19,635 | 32,125 | 21,578 | 19,598 | 34,663 |
| Rural | | | | | | |
| Attica | 13,694 | 10,394 | 13,509 | 13,793 | 11,700 | 17,353 |
| Crete | 39,104 | 28,559 | 37,277 | 39,847 | 28,915 | 42,531 |
| Eastern Macedonia & Thrace | 38,961 | 26,422 | 41,537 | 34,401 | 27,677 | 49,605 |
| Central Macedonia | 64,705 | 52,161 | 73,683 | 66,077 | 55,180 | 89,276 |
| Western Macedonia | 16,563 | 14,913 | 22,668 | 16,528 | 14,890 | 24,922 |
| Epirus | 23,151 | 19,373 | 34,634 | 24,574 | 19,204 | 38,581 |
| Thessaly | 28,666 | 23,314 | 37,423 | 28,471 | 23,633 | 43,065 |
| Western Greece | 39,925 | 29,645 | 44,082 | 38,463 | 29,605 | 50,372 |
| Central Greece | 41,112 | 33,323 | 49,337 | 36,763 | 31,450 | 56,374 |
| Peloponnese | 42,110 | 35,481 | 58,050 | 38,991 | 35,414 | 62,637 |

Table 10. Total smokers by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| Attica | 188,986 | 166,718 | 123,064 | 162,951 | 167,840 | 110,065 |
| Crete | 17,537 | 14,820 | 11,130 | 15,353 | 13,463 | 8,890 |
| Eastern Macedonia & Thrace | 3,836 | 3,055 | 2,641 | 2,872 | 2,840 | 2,168 |
| Central Macedonia | 50,578 | 47,110 | 38,496 | 44,442 | 44,773 | 32,730 |
| Western Macedonia | 0 | 0 | 0 | 0 | 0 | 0 |
| Epirus | 6,055 | 5,625 | 6,631 | 5,741 | 5,162 | 5,499 |
| Thessaly | 20,255 | 19,287 | 17,175 | 17,103 | 17,389 | 13,639 |
| Western Greece | 15,132 | 13,091 | 10,961 | 12,444 | 11,669 | 8,696 |
| Central Greece | 3,784 | 3,493 | 3,130 | 2,949 | 2,994 | 2,558 |
| Peloponnese | 3,166 | 3,255 | 2,619 | 2,407 | 2,800 | 1,868 |
| Intermediate | | | | | | |
| Attica | 62,377 | 55,659 | 39,651 | 53,220 | 55,544 | 34,980 |
| Crete | 8,050 | 6,883 | 4,988 | 6,976 | 6,198 | 3,929 |
| Eastern Macedonia & Thrace | 17,315 | 13,950 | 11,647 | 12,836 | 12,852 | 9,442 |
| Central Macedonia | 40,461 | 38,125 | 30,055 | 35,190 | 35,920 | 25,190 |
| Western Macedonia | 15,150 | 14,183 | 18,176 | 14,454 | 13,763 | 17,255 |
| Epirus | 5,179 | 4,862 | 5,532 | 4,861 | 4,427 | 4,508 |
| Thessaly | 9,219 | 8,882 | 7,640 | 7,707 | 7,936 | 5,988 |
| Western Greece | 10,371 | 9,077 | 7,338 | 8,445 | 8,021 | 5,740 |
| Central Greece | 14,564 | 13,600 | 11,752 | 11,236 | 11,556 | 9,459 |
| Peloponnese | 7,075 | 7,351 | 5,741 | 5,334 | 6,273 | 4,056 |
| Rural | | | | | | |
| Attica | 5,269 | 4,802 | 3,215 | 4,418 | 4,717 | 2,773 |
| Crete | 15,544 | 13,574 | 9,237 | 13,229 | 12,029 | 7,107 |
| Eastern Macedonia & Thrace | 13,777 | 11,332 | 8,910 | 10,038 | 10,279 | 7,074 |
| Central Macedonia | 26,063 | 25,079 | 18,561 | 22,255 | 23,253 | 15,195 |
| Western Macedonia | 13,651 | 12,907 | 15,881 | 12,880 | 12,433 | 14,647 |
| Epirus | 12,381 | 11,858 | 12,628 | 11,402 | 10,635 | 9,992 |
| Thessaly | 10,389 | 10,219 | 8,270 | 8,536 | 8,988 | 6,348 |
| Western Greece | 15,040 | 13,441 | 10,214 | 12,027 | 11,688 | 7,818 |
| Central Greece | 18,402 | 17,548 | 14,209 | 13,930 | 14,675 | 11,140 |
| Peloponnese | 10,532 | 11,145 | 8,284 | 7,829 | 9,378 | 5,769 |

# Hungary

Table 11. Total population by degree of urbanization and age-sex group.

| | Men | | | Women | | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| Central Hungary | 288,755 | 185,594 | 233,102 | 291,121 | 190,681 | 342,176 |
| Central Transdanubia | 16,706 | 11,334 | 14,699 | 15,562 | 11,186 | 20,340 |
| Western Transdanubia | 35,954 | 25,120 | 32,804 | 34,009 | 24,659 | 45,096 |
| Southern Transdanubia | 23,303 | 16,588 | 23,120 | 22,213 | 16,857 | 32,528 |
| Northern Hungary | 27,555 | 18,736 | 24,429 | 25,556 | 18,919 | 36,076 |
| Northern Great Plain | 55,455 | 36,449 | 45,098 | 52,183 | 36,630 | 63,669 |
| Southern Great Plain | 46,985 | 32,212 | 44,382 | 44,331 | 32,538 | 62,914 |
| Intermediate | | | | | | |
| Central Hungary | 144,860 | 93,107 | 116,941 | 146,047 | 95,659 | 171,660 |
| Central Transdanubia | 71,697 | 48,641 | 63,084 | 66,789 | 48,010 | 87,296 |
| Western Transdanubia | 53,580 | 37,434 | 48,886 | 50,681 | 36,748 | 67,204 |
| Southern Transdanubia | 42,802 | 30,469 | 42,465 | 40,800 | 30,962 | 59,746 |
| Northern Hungary | 63,710 | 43,319 | 56,481 | 59,088 | 43,742 | 83,411 |
| Northern Great Plain | 77,189 | 50,734 | 62,773 | 72,634 | 50,985 | 88,622 |
| Southern Great Plain | 67,112 | 46,011 | 63,394 | 63,321 | 46,476 | 89,864 |
| Rural | | | | | | |
| Central Hungary | 31,718 | 20,387 | 25,605 | 31,978 | 20,945 | 37,586 |
| Central Transdanubia | 75,455 | 51,191 | 66,390 | 70,289 | 50,526 | 91,872 |
| Western Transdanubia | 59,788 | 41,772 | 54,550 | 56,553 | 41,006 | 74,991 |
| Southern Transdanubia | 64,871 | 46,179 | 64,361 | 61,837 | 46,926 | 90,552 |
| Northern Hungary | 81,714 | 55,560 | 72,443 | 75,785 | 56,103 | 106,982 |
| Northern Great Plain | 97,233 | 63,909 | 79,074 | 91,496 | 64,225 | 111,635 |
| Southern Great Plain | 74,643 | 51,174 | 70,508 | 70,427 | 51,692 | 99,949 |

Table 12. Total smokers by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|-----------------------|---------|--------|--------|--------|--------|--------|
| Region | 18–39 | 40-54 | ≥55 | 18–39 | 40-54 | ≥55 |
| Urban | | | | | | |
| Central Hungary | 114,636 | 65,329 | 49,627 | 63,726 | 57,166 | 36,100 |
| Central Transdanubia | 9,324 | 5,783 | 5,021 | 5,440 | 5,044 | 3,753 |
| Western Transdanubia | 16,082 | 10,056 | 8,185 | 8,713 | 8,502 | 5,709 |
| Southern Transdanubia | 10,158 | 6,458 | 5,570 | 5,498 | 5,637 | 3,955 |
| Northern Hungary | 13,530 | 8,302 | 6,933 | 7,437 | 7,291 | 5,314 |
| Northern Great Plain | 25,204 | 14,846 | 11,500 | 13,662 | 12,868 | 8,271 |
| Southern Great Plain | 18,465 | 11,213 | 9,325 | 9,575 | 9,638 | 6,537 |
| Intermediate | | | | | | |
| Central Hungary | 63,811 | 36,656 | 28,569 | 36,658 | 32,381 | 21,217 |
| Central Transdanubia | 43,133 | 26,981 | 24,149 | 26,128 | 23,784 | 18,585 |
| Western Transdanubia | 26,351 | 16,617 | 13,903 | 14,784 | 14,188 | 9,926 |
| Southern Transdanubia | 20,554 | 13,175 | 11,682 | 11,514 | 11,617 | 8,484 |
| Northern Hungary | 34,117 | 21,118 | 18,153 | 19,452 | 18,743 | 14,280 |
| Northern Great Plain | 38,517 | 22,881 | 18,223 | 21,623 | 20,037 | 13,417 |
| Southern Great Plain | 29,281 | 17,930 | 15,291 | 15,691 | 15,560 | 10,945 |
| Rural | | | | | | |
| Central Hungary | 13,027 | 7,443 | 5,700 | 7,317 | 6,531 | 4,172 |
| Central Transdanubia | 43,168 | 26,845 | 23,535 | 25,487 | 23,495 | 17,750 |
| Western Transdanubia | 27,586 | 17,298 | 14,199 | 15,111 | 14,668 | 9,974 |
| Southern Transdanubia | 29,185 | 18,606 | 16,187 | 15,966 | 16,288 | 11,573 |
| Northern Hungary | 41,282 | 25,402 | 21,407 | 22,955 | 22,385 | 16,539 |
| Northern Great Plain | 45,563 | 26,912 | 21,026 | 24,969 | 23,404 | 15,227 |
| Southern Great Plain | 30,357 | 18,484 | 15,491 | 15,902 | 15,931 | 10,924 |

## **Poland**

Table 13. Total population by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| Łódzkie | 191,259 | 114,296 | 162,808 | 182,873 | 116,981 | 230,158 |
| Mazowieckie | 424,749 | 242,973 | 330,065 | 422,853 | 246,532 | 452,401 |
| Malopolskie | 216,365 | 123,945 | 155,542 | 211,271 | 123,750 | 204,558 |
| Śląskie | 452,539 | 279,143 | 382,154 | 436,539 | 281,496 | 504,044 |
| Lubelskie | 107,420 | 61,659 | 81,845 | 100,674 | 60,948 | 111,518 |
| Podkarpackie | 68,477 | 39,402 | 48,399 | 64,907 | 38,556 | 62,801 |
| Świętokrzyskie | 50,053 | 29,532 | 42,161 | 46,624 | 28,740 | 54,878 |
| Podlaskie | 85,219 | 51,125 | 64,784 | 79,722 | 50,298 | 85,952 |
| Wielkopolskie | 204,836 | 114,709 | 146,755 | 197,924 | 115,154 | 192,484 |
| Zachodniopomorskie | 100,956 | 58,876 | 82,373 | 96,300 | 57,989 | 106,584 |
| Lubuskie | 43,270 | 24,639 | 33,217 | 41,344 | 24,272 | 43,276 |
| Dolnośląskie | 215,571 | 122,836 | 176,115 | 208,635 | 122,628 | 237,598 |
| Opolskie | 21,056 | 13,344 | 17,541 | 20,251 | 13,134 | 23,160 |
| Kujawsko-Pomorskie | 149,704 | 87,405 | 115,224 | 144,422 | 88,344 | 152,026 |
| Warmińsko-Mazurskie | 69,743 | 40,544 | 50,286 | 65,706 | 39,743 | 65,737 |
| Pomorskie | 175,132 | 99,814 | 130,602 | 170,870 | 99,044 | 167,525 |
| Intermediate | , | , | , | , | , | , |
| Łódzkie | 83,269 | 49,761 | 70,882 | 79,618 | 50,930 | 100,205 |
| Mazowieckie | 216,245 | 123,700 | 168,040 | 215,279 | 125,512 | 230,322 |
| Malopolskie | 182,378 | 104,476 | 131,110 | 178,084 | 104,312 | 172,426 |
| Śląskie | 193,186 | 119,164 | 163,139 | 186,356 | 120,169 | 215,173 |
| Lubelskie | 78,329 | 44,961 | 59,680 | 73,410 | 44,442 | 81,317 |
| Podkarpackie | 136,577 | 78,586 | 96,530 | 129,457 | 76,899 | 125,255 |
| Świętokrzyskie | 42,249 | 24,927 | 35,587 | 39,354 | 24,259 | 46,321 |
| Podlaskie | 32,612 | 19,565 | 24,792 | 30,508 | 19,248 | 32,892 |
| Wielkopolskie | 130,247 | 72,939 | 93,316 | 125,852 | 73,222 | 122,394 |
| Zachodniopomorskie | 42,322 | 24,681 | 34,532 | 40,370 | 24,310 | 44,681 |
| Lubuskie | 37,758 | 21,500 | 28,985 | 36,077 | 21,180 | 37,763 |
| Dolnośląskie | 95,569 | 54,457 | 78,077 | 92,494 | 54,365 | 105,335 |
| Opolskie | 36,477 | 23,118 | 30,388 | 35,081 | 22,754 | 40,121 |
| Kujawsko-Pomorskie | 43,488 | 25,391 | 33,472 | 41,954 | 25,663 | 44,163 |
| Warmińsko-Mazurskie | 50,802 | 29,533 | 36,630 | 47,862 | 28,950 | 47,884 |
| Pomorskie | 88,601 | 50,497 | 66,072 | 86,444 | 50,107 | 84,752 |
| Rural | 00,001 | 00,101 | 00,012 | 00,111 | 00,101 | 01,102 |
| Łódzkie | 121,996 | 72,905 | 103,849 | 116,647 | 74,617 | 146,808 |
| Mazowieckie | 225,751 | 129,139 | 175,427 | 224,744 | 131,030 | 240,448 |
| Malopolskie | 163,112 | 93,440 | 117,260 | 159,272 | 93,292 | 154,212 |
| Śląskie | 84,623 | 52,198 | 71,461 | 81,631 | 52,638 | 94,254 |
| Lubelskie | 171,083 | 98,202 | 130,350 | 160,339 | 97,068 | 177,609 |
| Podkarpackie | 153,588 | 88,375 | 108,553 | 145,581 | 86,477 | 140,856 |
| Świętokrzyskie | 113,230 | 66,806 | 95,376 | 105,472 | 65,015 | 124,145 |

Table 13. (Continued)

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40-54 | ≥55 |
| Podlaskie | 77,339 | 46,398 | 58,794 | 72,350 | 45,647 | 78,005 |
| Wielkopolskie | 251,793 | 141,005 | 180,398 | 243,296 | 141,552 | 236,610 |
| Zachodniopomorskie | 136,157 | 79,405 | 111,095 | 129,878 | 78,208 | 143,748 |
| Lubuskie | 88,469 | 50,376 | 67,915 | 84,531 | 49,627 | 88,481 |
| Dolnośląskie | 163,354 | 93,082 | 133,456 | 158,098 | 92,924 | 180,046 |
| Opolskie | 97,286 | 61,656 | 81,047 | 93,564 | 60,685 | 107,006 |
| Kujawsko-Pomorskie | 149,283 | 87,159 | 114,900 | 144,015 | 88,095 | 151,598 |
| Warmińsko-Mazurskie | 121,430 | 70,592 | 87,555 | 114,401 | 69,198 | 114,456 |
| Pomorskie | 115,945 | 66,081 | 86,464 | 113,123 | 65,571 | 110,909 |

Table 14. Total smokers by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40-54 | ≥55 |
| Urban | | | | | | |
| Łódzkie | 60,859 | 54,405 | 45,684 | 54,332 | 30,614 | 45,318 |
| Mazowieckie | 148,322 | 124,135 | 102,188 | 138,315 | 71,371 | 99,483 |
| Malopolskie | 36,717 | 24,554 | 22,694 | 33,022 | 16,632 | 19,842 |
| Śląskie | 152,596 | 138,902 | 113,997 | 137,728 | 78,453 | 106,303 |
| Lubelskie | 35,814 | 30,423 | 24,128 | 31,400 | 30,072 | 23,207 |
| Podkarpackie | 24,255 | 20,347 | 15,212 | 21,549 | 11,335 | 14,049 |
| Świętokrzyskie | 13,549 | 12,389 | 9,984 | 11,735 | 6,320 | 8,956 |
| Podlaskie | 34,582 | 29,177 | 23,536 | 30,470 | 17,177 | 22,691 |
| Wielkopolskie | 60,365 | 51,458 | 37,980 | 54,350 | 27,741 | 34,647 |
| Zachodniopomorskie | 27,420 | 24,763 | 19,572 | 24,316 | 12,798 | 17,458 |
| Lubuskie | 27,213 | 18,908 | 19,468 | 25,038 | 13,658 | 20,383 |
| Dolnośląskie | 59,692 | 52,463 | 42,708 | 53,744 | 27,628 | 39,798 |
| Opolskie | 4,763 | 4,840 | 3,443 | 4,241 | 2,386 | 3,083 |
| Kujawsko-Pomorskie | 49,462 | 42,820 | 33,645 | 44,612 | 24,083 | 31,302 |
| Warmińsko-Mazurskie | 13,126 | 12,605 | 8,161 | 11,400 | 5,950 | 7,132 |
| Pomorskie | 29,545 | 28,277 | 18,937 | 26,553 | 13,232 | 16,149 |
| Intermediate | | | | | | |
| Łódzkie | 27,021 | 24,049 | 20,308 | 24,148 | 13,614 | 20,191 |
| Mazowieckie | 76,962 | 64,101 | 53,084 | 71,817 | 37,101 | 51,822 |
| Malopolskie | 31,716 | 30,371 | 19,614 | 28,529 | 14,374 | 17,174 |
| Śląskie | 66,417 | 60,166 | 49,676 | 59,988 | 34,200 | 46,434 |
| Lubelskie | 26,624 | 22,512 | 17,958 | 23,359 | 12,497 | 17,321 |
| Podkarpackie | 49,291 | 41,155 | 30,948 | 43,821 | 23,077 | 28,658 |
| Świętokrzyskie | 11,682 | 10,634 | 8,616 | 10,122 | 5,458 | 7,745 |
| Podlaskie | 13,462 | 11,305 | 9,176 | 11,871 | 6,700 | 8,874 |
| Wielkopolskie | 39,178 | 33,246 | 24,682 | 35,301 | 18,035 | 22,569 |
| Zachodniopomorskie | 11,740 | 10,556 | 8,388 | 10,419 | 5,487 | 7,497 |
| Lubuskie | 23,999 | 16,609 | 17,194 | 22,097 | 12,070 | 18,058 |
| Dolnośląskie | 27,027 | 23,651 | 19,355 | 24,344 | 12,531 | 18,075 |
| Opolskie | 8,437 | 8,540 | 6,108 | 7,518 | 4,232 | 5,477 |
| Kujawsko-Pomorskie | 14,651 | 12,624 | 9,975 | 13,224 | 7,145 | 9,305 |
| Warmińsko-Mazurskie | 9,790 | 9,368 | 6,092 | 8,510 | 4,441 | 5,334 |
| Pomorskie | 15,319 | 14,604 | 9,825 | 13,762 | 6,865 | 8,382 |
| Rural | | | | | | |
| Łódzkie | 42,455 | 37,152 | 32,037 | 38,027 | 21,520 | 32,151 |
| Mazowieckie | 85,853 | 70,303 | 59,470 | 80,324 | 41,654 | 58,621 |
| Malopolskie | 30,910 | 29,228 | 19,172 | 27,841 | 14,068 | 16,871 |
| Śląskie | 31,133 | 27,728 | 23,382 | 28,179 | 16,134 | 22,074 |
| Lubelskie | 62,257 | 51,752 | 42,168 | 54,740 | 29,402 | 41,045 |
| Podkarpackie | 59,208 | 48,589 | 37,342 | 52,759 | 27,906 | 34,918 |
| Świętokrzyskie | 33,754 | 30,230 | 24,979 | 29,300 | 15,851 | 22,644 |
| Podlaskie | 33,921 | 27,992 | 23,224 | 29,982 | 16,999 | 22,699 |
| Wielkopolskie | 81,430 | 67,964 | 51,486 | 73,524 | 37,695 | 47,488 |

Table 14. (Continued)

| | | Men | | Women | | |
|---------------------|--------|--------|--------|--------|--------|--------|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Zachodniopomorskie | 40,711 | 36,018 | 29,196 | 36,197 | 19,137 | 26,320 |
| Lubuskie | 58,363 | 39,822 | 41,992 | 53,863 | 29,553 | 44,639 |
| Dolnośląskie | 49,758 | 42,846 | 35,766 | 44,916 | 23,203 | 33,687 |
| Opolskie | 24,380 | 24,311 | 17,701 | 21,754 | 12,289 | 15,987 |
| Kujawsko-Pomorskie | 53,861 | 45,628 | 36,825 | 48,720 | 26,428 | 34,670 |
| Warmińsko-Mazurskie | 25,452 | 24,030 | 15,882 | 22,159 | 11,598 | 13,998 |
| Pomorskie | 21,844 | 20,571 | 14,050 | 19,661 | 9,829 | 12,056 |

## Romania

Table 15. Total population by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|--------------|---------|---------|---------|---------|---------|---------|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| North-West | 118,494 | 78,468 | 93,874 | 112,803 | 76,075 | 123,288 |
| Central | 105,047 | 71,537 | 91,367 | 98,015 | 69,435 | 116,693 |
| North-East | 136,912 | 95,862 | 119,840 | 124,116 | 87,857 | 152,514 |
| South-East | 126,652 | 96,245 | 124,266 | 116,364 | 91,508 | 159,515 |
| South | 92,679 | 71,780 | 89,519 | 84,251 | 67,073 | 118,306 |
| Bucharest | 331,228 | 191,549 | 227,613 | 345,974 | 208,623 | 325,318 |
| South-West | 83,607 | 65,845 | 82,889 | 77,011 | 62,128 | 106,055 |
| West | 84,314 | 58,920 | 71,332 | 79,981 | 57,447 | 94,264 |
| Intermediate | | | | | | |
| North-West | 100,605 | 66,622 | 79,702 | 95,773 | 64,590 | 104,675 |
| Central | 104,799 | 71,368 | 91,151 | 97,784 | 69,272 | 116,418 |
| North-East | 110,249 | 77,194 | 96,502 | 99,945 | 70,747 | 122,813 |
| South-East | 85,783 | 65,188 | 84,167 | 78,815 | 61,980 | 108,042 |
| South | 122,932 | 95,211 | 118,740 | 111,752 | 88,967 | 156,925 |
| Bucharest | 44,569 | 25,774 | 30,627 | 46,553 | 28,072 | 43,774 |
| South-West | 35,147 | 27,680 | 34,845 | 32,374 | 26,118 | 44,583 |
| West | 87,578 | 61,201 | 74,093 | 83,077 | 59,670 | 97,913 |
| Rural | | | | | | |
| North-West | 192,525 | 127,493 | 152,524 | 183,279 | 123,604 | 200,314 |
| Central | 150,261 | 102,328 | 130,693 | 140,204 | 99,322 | 166,921 |
| North-East | 240,326 | 168,270 | 210,358 | 217,865 | 154,217 | 267,713 |
| South-East | 145,494 | 110,563 | 142,753 | 133,676 | 105,122 | 183,246 |
| South | 227,014 | 175,824 | 219,274 | 206,369 | 164,293 | 289,788 |
| Bucharest | 13,727 | 7,938 | 9,433 | 14,338 | 8,646 | 13,482 |
| South-West | 171,627 | 135,166 | 170,153 | 158,086 | 127,535 | 217,706 |
| West | 111,413 | 77,857 | 94,259 | 105,688 | 75,911 | 124,562 |

Table 16. Total smokers by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|--------------|---------|--------|--------|---------|--------|--------|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40-54 | ≥55 |
| Urban | | | | | | |
| North-West | 52,232 | 29,504 | 11,058 | 35,070 | 18,722 | 10,356 |
| Central | 55,234 | 32,821 | 14,454 | 38,059 | 21,858 | 13,326 |
| North-East | 56,202 | 33,302 | 12,655 | 35,385 | 19,671 | 11,423 |
| South-East | 58,133 | 37,863 | 15,620 | 38,039 | 23,801 | 14,324 |
| South | 60,149 | 42,042 | 21,359 | 43,330 | 29,096 | 20,940 |
| Bucharest | 175,816 | 88,821 | 36,623 | 136,002 | 66,572 | 37,834 |
| South-West | 62,981 | 46,098 | 28,265 | 48,994 | 34,705 | 27,797 |
| West | 55,082 | 34,775 | 17,262 | 41,502 | 25,185 | 16,939 |
| Intermediate | | | | | | |
| North-West | 30,222 | 16,462 | 5,404 | 18,896 | 9,753 | 4,983 |
| Central | 39,467 | 22,545 | 8,468 | 25,130 | 13,868 | 7,637 |
| North-East | 30,329 | 17,361 | 5,829 | 17,840 | 9,615 | 5,195 |
| South-East | 27,116 | 17,021 | 6,111 | 16,488 | 9,960 | 5,510 |
| South | 61,700 | 41,426 | 17,324 | 40,879 | 26,201 | 16,461 |
| Bucharest | 16,994 | 8,255 | 2,897 | 12,141 | 5,710 | 2,928 |
| South-West | 21,953 | 15,498 | 7,666 | 15,795 | 10,659 | 7,227 |
| West | 44,367 | 26,910 | 10,981 | 30,755 | 17,806 | 10,438 |
| Rural | | | | | | |
| North-West | 59,028 | 32,205 | 10,631 | 37,022 | 19,134 | 9,795 |
| Central | 57,625 | 32,980 | 12,468 | 36,818 | 20,351 | 11,267 |
| North-East | 67,532 | 38,702 | 13,063 | 39,826 | 21,482 | 11,646 |
| South-East | 46,922 | 29,498 | 10,649 | 28,620 | 17,314 | 9,602 |
| South | 115,596 | 77,767 | 32,781 | 76,893 | 49,386 | 31,210 |
| Bucharest | 5,329 | 2,593 | 916 | 3,821 | 1,800 | 926 |
| South-West | 108,365 | 76,639 | 38,284 | 78,284 | 52,953 | 36,161 |
| West | 57,255 | 34,794 | 14,318 | 39,844 | 23,122 | 13,640 |

# Spain

Table 17. Total population by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| Galicia | 139,534 | 121,795 | 176,058 | 136,440 | 123,324 | 218,339 |
| Asturias | 72,644 | 69,132 | 100,039 | 70,868 | 70,372 | 128,027 |
| Cantabria | 24,397 | 21,800 | 27,802 | 23,570 | 21,561 | 33,951 |
| Basque Country | 88,940 | 85,404 | 110,728 | 87,237 | 85,114 | 136,908 |
| Rioja | 21,075 | 18,677 | 23,520 | 20,680 | 17,950 | 27,082 |
| Aragon | 94,717 | 82,984 | 105,097 | 89,549 | 78,381 | 123,905 |
| Madrid | 750,580 | 621,299 | 643,682 | 765,922 | 646,188 | 836,540 |
| Castile-Leon | 123,946 | 114,994 | 167,830 | 117,132 | 110,681 | 193,523 |
| Castile-La Mancha | 77,033 | 61,481 | 70,026 | 71,545 | 57,364 | 79,358 |
| Extremadura | 37,913 | 31,315 | 38,638 | 35,897 | 30,018 | 44,588 |
| Cataluna | 622,139 | 528,437 | 603,330 | 616,187 | 514,711 | 738,443 |
| Valencia | 250,809 | 212,258 | 245,849 | 241,774 | 205,700 | 291,282 |
| Baleares | 67,560 | 53,211 | 52,684 | 65,876 | 50,186 | 60,275 |
| Andalucia | 514,380 | 403,975 | 430,155 | 497,197 | 399,287 | 509,349 |
| Murcia | 106,587 | 81,749 | 80,138 | 100,255 | 76,955 | 93,640 |
| Intermediate | | | | | | |
| Galicia | 85,953 | 75,026 | 108,452 | 84,048 | 75,968 | 134,497 |
| Asturias | 22,800 | 21,698 | 31,399 | 22,243 | 22,087 | 40,183 |
| Cantabria | 36,155 | 32,306 | 41,202 | 34,929 | 31,953 | 50,314 |
| Basque Country | 63,163 | 60,652 | 78,637 | 61,954 | 60,446 | 97,230 |
| Rioja | 10,961 | 9,714 | 12,233 | 10,756 | 9,336 | 14,086 |
| Aragon | 32,202 | 28,213 | 35,731 | 30,445 | 26,648 | 42,125 |
| Madrid | 112,184 | 92,861 | 96,207 | 114,477 | 96,581 | 125,032 |
| Castile-Leon | 65,343 | 60,624 | 88,479 | 61,751 | 58,350 | 102,023 |
| Castile-La Mancha | 31,445 | 25,097 | 28,585 | 29,205 | 23,416 | 32,394 |
| Extremadura | 12,674 | 10,468 | 12,916 | 12,000 | 10,035 | 14,905 |
| Cataluna | 295,469 | 250,967 | 286,536 | 292,642 | 244,449 | 350,704 |
| Valencia | 322,744 | 273,137 | 316,362 | 311,118 | 264,697 | 374,826 |
| Baleares | 37,489 | 29,527 | 29,235 | 36,555 | 27,848 | 33,446 |
| Andalucia | 273,472 | 214,775 | 228,694 | 264,337 | 212,283 | 270,797 |
| Murcia | 38,747 | 29,718 | 29,132 | 36,445 | 27,975 | 34,041 |
| Rural | | | | | | |
| Galicia | 131,903 | 115,134 | 166,430 | 128,978 | 116,579 | 206,398 |
| Asturias | 34,172 | 32,520 | 47,059 | 33,337 | 33,103 | 60,225 |
| Cantabria | 17,752 | 15,862 | 20,230 | 17,150 | 15,688 | 24,704 |
| Basque Country | 117,805 | 113,122 | 146,665 | 115,550 | 112,738 | 181,342 |
| Rioja | 10,146 | 8,992 | 11,323 | 9,956 | 8,642 | 13,038 |
| Aragon | 54,760 | 47,977 | 60,761 | 51,772 | 45,315 | 71,635 |
| Madrid | 51,974 | 43,022 | 44,572 | 53,036 | 44,745 | 57,926 |
| Castile-Leon | 127,454 | 118,250 | 172,581 | 120,448 | 113,814 | 199,001 |
| Castile-La Mancha | 202,103 | 161,300 | 183,719 | 187,706 | 150,499 | 208,203 |

Table 17. (Continued)

| | | Men | | Women | | |
|-------------|---------|---------|---------|---------|---------|---------|
| Region | 18–39 | 40-54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Extremadura | 106,404 | 87,886 | 108,437 | 100,746 | 84,247 | 125,137 |
| Cataluna | 114,137 | 96,946 | 110,686 | 113,045 | 94,428 | 135,474 |
| Valencia | 127,367 | 107,790 | 124,848 | 122,779 | 104,459 | 147,920 |
| Baleares | 72,665 | 57,231 | 56,665 | 70,854 | 53,978 | 64,829 |
| Andalucia | 474,169 | 372,395 | 396,528 | 458,329 | 368,074 | 469,531 |
| Murcia | 83,518 | 64,056 | 62,794 | 78,556 | 60,300 | 73,373 |

Table 18. Total smokers by degree of urbanization and age-sex group.

| | | Men | | | Women | |
|---|---|---|---|---|---|---|
| Region | 18–39 | 40–54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Urban | | | | | | |
| Galicia | 61,269 | 63,589 | 43,979 | 55,272 | 42,793 | 30,982 |
| Asturias | 38,814 | 42,558 | 32,813 | 35,399 | 30,809 | 24,978 |
| Cantabria | 11,874 | 12,401 | 8,032 | 10,661 | 8,461 | 5,721 |
| Basque Country | 30,008 | 35,477 | 19,710 | 26,773 | 21,857 | 13,294 |
| Rioja | 8,525 | 9,090 | 5,273 | 7,681 | 5,663 | 3,399 |
| Aragon | 38,313 | 40,388 | 23,563 | 33,258 | 24,729 | 15,550 |
| Madrid | 297,155 | 296,795 | 140,323 | 278,030 | 198,897 | 101,723 |
| Castile-Leon | 56,358 | 61,855 | 43,938 | 49,242 | 40,000 | 28,990 |
| Castile-La Mancha | 36,668 | 34,368 | 19,516 | 31,580 | 21,879 | 12,777 |
| Extremadura | 17,713 | 17,233 | 10,498 | 15,533 | 11,200 | 6,969 |
| Cataluna | 189,068 | 200,066 | 94,481 | 169,575 | 117,663 | 62,325 |
| Valencia | 103,985 | 105,513 | 56,914 | 92,164 | 66,770 | 37,896 |
| Baleares | 20,106 | 19,773 | 8,045 | 17,740 | 11,207 | 4,949 |
| Andalucia | 226,224 | 211,239 | 107,711 | 201,763 | 138,792 | 72,480 |
| Murcia | 33,362 | 31,776 | 13,006 | 28,452 | 18,169 | 8,222 |
| Intermediate | | | | | | |
| Galicia | 36,728 | 38,278 | 26,126 | 33,081 | 25,540 | 18,318 |
| Asturias | 11,911 | 13,110 | 9,969 | 10,843 | 9,409 | 7,542 |
| Cantabria | 17,168 | 18,001 | 11,504 | 15,388 | 12,177 | 8,148 |
| Basque Country | 20,635 | 24,491 | 13,455 | 18,388 | 14,979 | 9,042 |
| Rioja | 4,308 | 4,611 | 2,641 | 3,875 | 2,850 | 1,695 |
| Aragon | 12,655 | 13,393 | 7,714 | 10,969 | 8,136 | 5,068 |
| Madrid | 43,135 | 43,245 | 20,194 | 40,296 | 28,752 | 14,579 |
| Castile-Leon | 28,940 | 31,882 | 22,359 | 25,244 | 20,446 | 14,671 |
| Castile-La Mancha | 14,590 | 13,733 | 7,695 | 12,546 | 8,666 | 5,008 |
| Extremadura | 5,770 | 5,636 | 3,388 | 5,052 | 3,632 | 2,237 |
| Cataluna | 86,809 | 92,205 | 43,095 | 77,755 | 53,828 | 28,337 |
| Valencia | 130,066 | 132,499 | 70,580 | 115,083 | 83,168 | 46,778 |
| Baleares | 10,786 | 10,642 | 4,286 | 9,501 | 5,990 | 2,629 |
| Andalucia | 117,073 | 109,729 | 55,230 | 104,228 | 71,497 | 36,964 |
| Murcia | 11,733 | 11,213 | 4,542 | 9,990 | 6,367 | 2,859 |
| Rural | | | | | | |
| Galicia | 51,706 | 54,539 | 35,816 | 46,342 | 35,487 | 24,747 |
| Asturias | 16,604 | 18,497 | 13,492 | 15,038 | 12,933 | 10,021 |
| Cantabria | 7,792 | 8,268 | 5,077 | 6,949 | 5,452 | 3,536 |
| Basque Country | 34,811 | 41,765 | 22,205 | 30,887 | 24,971 | 14,761 |
| Rioja | 3,640 | 3,943 | 2,176 | 3,259 | 2,378 | 1,378 |
| Aragon | 19,648 | 21,038 | 11,678 | 16,950 | 12,471 | 7,572 |
| Madrid | 18,217 | 18,482 | 8,322 | 16,945 | 11,996 | 5,926 |
| Castile-Leon | 51,899 | 57,883 | 39,021 | 45,048 | 36,181 | 25,213 |
| Castile-La Mancha | 86,500 | 82,392 | 44,350 | 73,994 | 50,688 | 28,420 |
| Extremadura | 44,626 | 44,119 | 25,483 | 38,868 | 27,709 | 16,568 |
| Cataluna | 30,189 | 32,399 | 14,688 | 26,927 | 18,527 | 9,564 |

Table 18. (Continued)

| | | Men | | Women | | |
|-----------|---------|---------|--------|---------|---------|--------|
| Region | 18–39 | 40-54 | ≥55 | 18–39 | 40–54 | ≥55 |
| Valencia | 46,922 | 48,376 | 24,820 | 41,327 | 29,625 | 16,227 |
| Baleares | 18,798 | 18,743 | 7,321 | 16,495 | 10,337 | 4,447 |
| Andalucia | 186,206 | 176,664 | 85,531 | 164,998 | 112,263 | 56,438 |
| Murcia | 22,784 | 22,016 | 8,640 | 19,325 | 12,235 | 5,386 |

# Summary statistics of the weights

The following tables show the means, standard deviations and coefficients of variation for the weights in the regions crossed with urbanization (following merging as indicated in Appendix A).

Table 19. Germany Wave 1 inflation weights: summary statistics.

| Region | | N | Sum | Mean | SD | CV |
|---|---|---|---|---|---|---|
| Baden-Württemberg | Urban | 37 | 445,212 | 12032.76 | 4447.40 | 36.96 |
| | Intermediate | 65 | 1,109,603 | 17070.82 | 6026.89 | 35.31 |
| | Rural | 29 | 331,851 | 11443.14 | 6248.86 | 54.61 |
| Bayern | Urban | 50 | 882,197 | 17643.94 | 12006.08 | 68.05 |
| | Intermediate | 70 | 1,005,773 | 14368.19 | 6577.90 | 45.78 |
| | Rural | 50 | 728,942 | 14578.84 | 4399.03 | 30.17 |
| Berlin | Urban | 30 | 1,033,241 | 34441.37 | 13104.80 | 38.05 |
| Former East Germany | Urban | 51 | 912,376 | 17889.73 | 5496.05 | 30.72 |
| | Intermediate | 58 | 991,376 | 17092.69 | 7876.08 | 46.08 |
| | Rural | 45 | 917,604 | 20391.20 | 11880.10 | 58.26 |
| Hamberg/Bremen/ | Urban | 96 | 1,359,424 | 14160.67 | 4740.62 | 33.48 |
| Schleswig-Holstein/ | Intermediate | 62 | 1,227,621 | 19800.34 | 8780.17 | 44.34 |
| Niedersachsen | Rural | 40 | 771,030 | 19275.75 | 9194.27 | 47.70 |
| Urban areas of Hessen* | Urban | 114 | 3,003,094 | 26342.93 | 10706.42 | 40.64 |
| Intermediate areas of Hessen <sup>†</sup> | Intermediate | 78 | 1,167,432 | 14967.08 | 7122.50 | 47.59 |
| Rest of Nordrhien-Westfalen | Intermediate | 78 | 1,636,560 | 20981.54 | 8773.90 | 41.82 |
| Rural ares of Hessen <sup>‡</sup> | Rural | 50 | 814,089 | 16281.78 | 5088.18 | 31.25 |

<sup>\*</sup>Urban areas of Hessen/Nordrhein-Westfalen/Rheinland-Pfalz

Table 20. Greece Wave 1 inflation weights: summary statistics.

| Region | | N | Sum | Mean | SD | CV |
|---|---|---|---|---|---|---|
| Attica | Urban | 400 | 1,246,249 | 3115.62 | 1144.37 | 36.73 |
| Crete | Urban | 50 | 188,937 | 3778.74 | 1635.62 | 43.28 |
| Northern Greece | Urban | 30 | 310,254 | 10341.80 | 4403.45 | 42.58 |
| | Intermediate | 180 | 405,333 | 2251.85 | 568.32 | 25.24 |
| | Rural | 100 | 343,111 | 3431.11 | 1336.80 | 38.96 |
| Central Greece | Urban | 50 | 211,864 | 4237.28 | 1501.49 | 35.44 |
| | Intermediate | 99 | 204,361 | 2064.25 | 1134.32 | 54.95 |
| | Rural | 91 | 265,819 | 2921.09 | 1374.57 | 47.06 |

<sup>†</sup>Intermediate areas of Hessen/Rheinland-Pfalz/Saarland

<sup>&</sup>lt;sup>‡</sup>Rural ares of Hessen/Nordrhein-Westfalen/Rheinland-Pfalz

Table 21. Hungary Wave 1 inflation weights: summary statistics.

| Region | | N | Sum | Mean | SD | CV |
|---|---|---|---|---|---|---|
| Central Hungary | Urban | 192 | 386,584 | 2013.46 | 1035.13 | 51.41 |
| | Intermediate | 109 | 263,482 | 2417.27 | 1240.71 | 51.33 |
| Urban Transdanubia* | Urban | 60 | 128,888 | 2148.13 | 949.29 | 44.19 |
| Rest of Central Transdanubia | Intermediate | 40 | 162,760 | 4069.00 | 3075.88 | 75.59 |
| | Rural | 40 | 160,280 | 4007.00 | 1841.17 | 45.95 |
| Rest of Western Transdanubia | Intermediate | 30 | 95,769 | 3192.30 | 1982.95 | 62.12 |
| | Rural | 50 | 98,836 | 1976.72 | 686.94 | 34.75 |
| Rest of Southern Transdanubia | Intermediate | 40 | 77,026 | 1925.65 | 592.38 | 30.76 |
| | Rural | 40 | 107,805 | 2695.13 | 1452.07 | 53.88 |
| Urban Nothern/Great Plain <sup>†</sup> | Urban | 90 | 199,911 | 2221.23 | 1128.61 | 50.81 |
| Rest of Northern Hungary | Intermediate | 50 | 125,863 | 2517.26 | 1109.38 | 44.07 |
| | Rural | 50 | 149,970 | 2999.40 | 1155.13 | 38.51 |
| Rest of Northern Great Plain | Intermediate | 60 | 134,698 | 2244.97 | 586.84 | 26.14 |
| | Rural | 50 | 157,101 | 3142.02 | 1773.08 | 56.43 |
| Rest of Southern Great Plain | Intermediate | 59 | 104,698 | 1774.54 | 560.43 | 31.58 |
| | Rural | 40 | 107,089 | 2677.23 | 812.45 | 30.35 |

<sup>\*</sup>Urban areas of Central/Western/Southern Transdanubia

<sup>&</sup>lt;sup>†</sup>Urban Northern Hungary and Northern & Southern Great Plain

Table 22. Poland Wave 1 inflation weights: summary statistics.

| Region | | N | Sum | Mean | SD | CV |
|---|---|---|---|---|---|---|
| Lodzkie (NUTS2) | Urban | 29 | 291,212 | 10041.79 | 5439.11 | 54.16 |
| | Intermediate | 22 | 129,331 | 5878.68 | 2756.69 | 46.89 |
| | Rural | 28 | 203,342 | 7262.21 | 3797.19 | 52.29 |
| Mazowieckie (NUTS2) | Urban | 64 | 683,814 | 10684.59 | 3694.32 | 34.58 |
| | Intermediate | 44 | 354,887 | 8065.61 | 2047.52 | 25.39 |
| | Rural | 48 | 396,225 | 8254.69 | 2376.85 | 28.79 |
| Poludniowy (NUTS1) | Urban | 75 | 881,440 | 11752.53 | 5379.99 | 45.78 |
| | Intermediate | 90 | 458,659 | 5096.21 | 2650.69 | 52.01 |
| | Rural | 63 | 286,720 | 4551.11 | 1933.68 | 42.49 |
| Wschondi (NUTS1) | Urban | 48 | 502,357 | 10465.77 | 5085.35 | 48.59 |
| | Intermediate | 41 | 452,866 | 11045.51 | 3563.82 | 32.26 |
| | Rural | 90 | 853,661 | 9485.12 | 5294.18 | 55.82 |
| Polnocno-Zachodni (NUTS1) | Urban | 53 | 517,536 | 9764.83 | 4614.77 | 47.26 |
| | Intermediate | 53 | 337,125 | 6360.85 | 3525.60 | 55.43 |
| | Rural | 52 | 815,398 | 15680.73 | 7643.61 | 48.75 |
| Poludniowo-Zachodni (NUTS1) | Urban | 21 | 298,789 | 14228.05 | 3551.69 | 24.96 |
| | Intermediate | 25 | 165,295 | 6611.80 | 2475.81 | 37.45 |
| | Rural | 18 | 346,598 | 19255.44 | 6465.94 | 33.58 |
| Polnocny (NUTS1) | Urban | 51 | 416,991 | 8176.29 | 5196.16 | 63.55 |
| | Intermediate | 34 | 179,216 | 5271.06 | 2790.68 | 52.94 |
| | Rural | 57 | 457,262 | 8022.14 | 5666.73 | 70.64 |

Table 23. Romania Wave 1 inflation weights: summary statistics.

| Region | | N | Sum | Mean | SD | CV |
|---|---|---|---|---|---|---|
| North-West + Central | Urban | 69 | 332,694 | 4821.65 | 1427.97 | 29.62 |
| | Intermediate | 70 | 202,835 | 2897.64 | 2036.15 | 70.27 |
| | Rural | 100 | 339,324 | 3393.24 | 1354.23 | 39.91 |
| North-East | Urban | 49 | 168,638 | 3441.59 | 1530.90 | 44.48 |
| | Intermediate | 60 | 168,375 | 2806.25 | 1349.84 | 48.10 |
| | Rural | 80 | 192,251 | 2403.14 | 1426.19 | 59.35 |
| South-East | Urban | 63 | 187,780 | 2980.63 | 1293.91 | 43.41 |
| | Rural | 51 | 142,605 | 2796.18 | 1826.73 | 65.33 |
| South + Bucharest | Urban | 120 | 758,584 | 6321.53 | 3952.70 | 62.53 |
| | Intermediate | 70 | 252,916 | 3613.09 | 2677.76 | 74.11 |
| | Rural | 80 | 399,018 | 4987.73 | 1794.99 | 35.99 |
| South-West + West | Urban | 59 | 439,585 | 7450.59 | 4145.60 | 55.64 |
| | Intermediate | 40 | 220,055 | 5501.38 | 2343.32 | 42.60 |
| | Rural | 90 | 573,659 | 6373.99 | 3651.28 | 57.28 |

Table 24. Spain Wave 1 inflation weights: summary statistics.

| Region | | N | Sum | Mean | SD | CV |
|---|---|---|---|---|---|---|
| Galicia/Asturias/ | Urban | 40 | 560,405 | 14010.12 | 6740.35 | 48.11 |
| Cantabria | Intermediate | 40 | 323,241 | 8081.03 | 3386.17 | 41.90 |
| | Rural | 30 | 372,296 | 12409.87 | 6325.76 | 50.97 |
| Pais Vasco/Rioja/ | Urban | 51 | 362,551 | 7108.84 | 3309.10 | 46.55 |
| Aragon | Intermediate | 30 | 178,905 | 5963.50 | 2078.56 | 34.85 |
| | Rural | 19 | 275,531 | 14501.63 | 6948.82 | 47.92 |
| Madrid/Leon/La Mancha/ | Urban | 160 | 1,829,240 | 11432.75 | 4960.97 | 43.39 |
| Extremadura | Intermediate | 60 | 421,696 | 7028.27 | 4243.97 | 60.38 |
| | Rural | 50 | 898,850 | 17977.00 | 11392.04 | 63.37 |
| Valencia/Baleares | Urban | 60 | 545,062 | 9084.37 | 4592.59 | 50.55 |
| | Intermediate | 60 | 622,008 | 10366.80 | 3414.61 | 32.94 |
| Cataluna/Valencia | Rural | 20 | 339,591 | 16979.55 | 3857.49 | 22.72 |
| Rest of Cataluna | Urban | 110 | 833,178 | 7574.35 | 2862.50 | 37.79 |
| | Intermediate | 50 | 382,029 | 7640.58 | 3163.80 | 41.41 |
| Andalucia/Murcia | Urban | 111 | 1,091,196 | 9830.59 | 4628.63 | 47.08 |
| | Intermediate | 80 | 541,425 | 6767.81 | 3206.79 | 47.38 |
| | Rural | 30 | 872,486 | 29082.87 | 11734.24 | 40.35 |

### D Field materials

Every Interviewer going into the field should have the following: Field preparatory materials:

- Interviewer's tablets (using NFIELD software in each country)
- ID card
- Survey manual and maps of the sampling points were loaded on the tablet
- Incentives

### Every Supervisor had the following field materials:

- Maps of selected survey areas, where possible.
- Additional interviewing tablet

## Survey information letter and consent

The following are the scripts used for both the information letter and consent:

### **Selected Respondent Information Letter:**

Research Project: International Tobacco Control 6 European Country Project (ITC 6E Project)

Human Research Ethics Committee, University of Waterloo: ORE # 21262, IRBs

#### What is this research about?

The International Tobacco Control (ITC) Project 6-European Country Study is a project under the European Regulatory Science on Tobacco: Policy implementation to reduce lung diseases (EUREST-PLUS). The objectives of EUREST-PLUS are to monitor and evaluate the impact of the tobacco control policies within the Tobacco Products Directive (TPD), the newly adopted legislation in the EU, and assess these within the context of the WHO Framework Convention on Tobacco Control (FCTC) ratification at a European level. The primary objective of the project is to evaluate the psychosocial and behavioural impact of the TPD. The aims of this research are to find out:

- 1. The impact of specific tobacco control policies within the TPD on residents of six European countries (Germany, Greece, Hungary, Poland, Romania, and Spain),
- 2. The prevalence and patterns of tobacco use behaviour within these countries,

3. The tobacco use behaviour and the impact of tobacco control policies between these countries and other countries within the ITC Project.

### Who is conducting this research?

The ITC 6E Project is led and coordinated by the ITC Project at the University of Waterloo (UW) in Canada in collaboration with European Network of Smoking and Tobacco Prevention (Belgium) and research partners from the 6 project countries. The overall international project is being led by Professor Geoffrey T. Fong from the University of Waterloo, Canada, in collaboration with Dr. Ute Mons, German Cancer Research Center; Prof. Yiannis Tountas, University of Athens; Prof. Witold Zatonski, Poland Health Promotion Foundation; Dr. Krzysztof Przewozniak, Poland Health Promotion Foundation; Prof. Antigona Trofor, Aer Pur Romania; Prof. Esteve Fernandez, Institut Català d'Oncologia; Dr. Tibor Demjén, Smoking or Health Hungarian Foundation; Prof. Aristidis Tsatsakis, University of Crete; and Mr. Nicolas Bécuwe, Kantar Public Brussels.

### What are we asking of you?

This research involves completing the survey interview (approximately 35 minutes) today. We plan to return approximately every 18 months to do follow-up surveys because we are interested in how peopleâAZs opinions and behaviours might change over time.

### **Survey Participation**

If you agree to participate in this research, first we will need to ask you a few essential questions for statistical purposes and to determine whether you are eligible. If you are not eligible, or if you do not answer these essential questions, we will not proceed further with the interview. If you are eligible, we will proceed with the interview, which will take about 35 minutes.

Participation is voluntary, and you may skip any non-essential questions if you wish. You may stop and start again if you cannot complete the survey all at one time. Once we are finished, a token of appreciation will be provided for your participation.

#### Risk

Participants will not face any risk or harm to their well-being either physically, psychologically, socially or culturally throughout completion of the survey.

#### **Possible Benefits**

This study will help the researchers to evaluate and understand the effects of national-level tobacco control policies in European Union Member States. Also policy makers throughout the world will be able to use this evidence to create and implement tobacco control policies for demonstrated effectiveness.

### **Confidentiality and Security of Data**

All the information you provide is treated as strictly confidential. Data from this research will not be destroyed, but any identifying information about you such as name and address will be removed so that your answers cannot be linked back to you.

The data will be held in secure electronic files at the survey firm TNS Opinion (Belgium) and at the University of Waterloo (Canada) on computers that have security certificates, are password protected, and can only be accessed by the research team. Eventually, after two years, the data without names or personal information may be shared with other health researchers.

If you wish to discuss any questions or concerns about this research project, please contact:

Dr. Constantine Vardavas, Principal Investigator, EUREST-PLUS, European Network on Smoking and Tobacco Prevention. Tel: \*\*\*\*\*\*\*\*\*.

OR

Dr. Geoffrey T. Fong, Principal Investigator, ITC Project, Department of Psychology, University of Waterloo, Canada. Tel: +1 519 888 4567 ext. 35811.

If you wish to lodge a complaint concerning the manner in which this research is being conducted, please contact:

[ethics contact]

If you feel that the local ethics committee has not resolved your concerns to your satisfaction, you may wish to contact the Human Research Ethics Committee in Canada that is overseeing the project:

Office of Research Ethics, University of Waterloo, 200 University Avenue West, Waterloo, Ontario, Canada N2L 3G1, Tel: + 1 519 888 4567 ext. 36005

### **BI49260**

#### Ask all.

Thank you. This is a comprehensive survey of smokers in this and other European Union member countries that has to do with beliefs, attitudes, knowledge, and behavior about tobacco use. It is being carried out by researchers from the EU and an international group.

This project is funded by an ongoing grant from the EU Horizon 2020. A major goal of the survey is to examine how smokers in this country differ or are the same in their views towards smoking.

We will talk to you for about 35 minutes, depending on your answers, and we think you will find the questions quite interesting. In addition, we will provide a token of appreciation for your involvement in this survey.

All personal information you provide is treated as strictly confidential, subject to legal requirements and limitations. It will be held in secure storage and password protected at TNS Opinion, Belgium and the University of Waterloo, Canada and only be accessed by this research team. Any identifying information about you will be removed before the data are securely stored, so that your answers cannot be linked back to you. After two years, the survey data, but not your name or other identifying information, will be shared with authorized researchers in other countries, as it will be used to make comparisons of smoking behaviour and attitudes across countries.

#### **BI49235**

### Ask all.

Would you be willing to answer the 35-minute survey today and then again in 12-18 months for a second token of our appreciation?

1 Yes

2 No

3 Time is not convenient

See HelpScreens for answers to any questions about follow-up surveys and contacts.

If response=1, go to FR225.

If response=2, go to BI439.

If response=3, make appointment and terminate.

### **BI49439**

#### Ask if BI235=2.

We understand how you feel. We really appreciate your participation. The difference between this and most other surveys is that this is an EU and international research project and we are talking to the same people a number of times to better understand what affects their opinions and smoking behaviour. This is why your participation is so important to us.

Can we just start with a few questions and see how it goes? (If hesitates, say) Or would another time be better?

1 Yes

2 No

3 Another time would be better

If response=1, go to FR225.

If response=2, go to BI901. (enter Indivdisp)

If response=3, make appointment and end interview.

| | T70 1 | 4 | |
|---|-------|----------|-------|
| H | Hinai | outcomes | ratec |
| 1 | rma | outcomes | Iaics |

Table 25. Final outcome rates

| | Germany | Greece | Hungary Poland | Poland | Romania | Snain |
|---|---|---|---|---|---|---|
| 1. Number of addresses approached/attempted | 10325 | 3537 | 2754 | 3421 | 4490 | 4114 |
| 2. Number of addresses where contact has been made | 8259 | 2856 | 2404 | 3028 | 2778 | 3853 |
| 3. Number of contacted addresses with eligibility determined | 3086 | 1295 | 1791 | 2154 | 2065 | 2451 |
| 4. Number of contacted addresses with no eligible respondents | 1982 | 466 | 972 | 1163 | 1134 | 1509 |
| 5. Number of contacted addresses with eligible respondents | 1104 | 829 | 819 | 991 | 931 | 942 |
| 6. Number of addresses with eligible respondents, members selected | 1085 | 823 | 809 | 976 | 911 | 936 |
| 7. Eligibility rate for households, given determination (5./3.) | 0.358 | 0.640 | 0.457 | 0.460 | 0.451 | 0.384 |
| 8. Estimated eligible households among attempted (7.*1.) | 3694 | 2264 | 1259 | 1574 | 2024 | 1581 |
| 9. Number of individuals selected for interview | 1425 | 1116 | 1078 | 1265 | 1254 | 1234 |
| 10. Number of individual refusals or break offs | 200 | 91 | 64 | 227 | 232 | 219 |
| 11. Number of completed interviews | 1003 | 1000 | 1000 | 1006 | 1003 | 1001 |
| Household contact rate (2./1.) | 0.800 | 0.807 | 0.873 | 0.885 | 0.619 | 0.937 |
| Household cooperation rate, given eligible (6./5.) | 0.983 | 0.993 | 0.988 | 0.985 | 0.979 | 0.994 |
| Household response rate (6./8.) | 0.294 | 0.363 | 0.642 | 0.620 | 0.450 | 0.592 |
| Individual cooperation rate (11./(11.+10.)) | 0.834 | 0.917 | 0.940 | 0.816 | 0.812 | 0.820 |
| Individual response rate, given selection (11./9.) | 0.704 | 0.896 | 0.928 | 0.795 | 0.800 | 0.811 |

## **G** Country profiles

#### **GERMANY**

Germany has an estimated population of 82 million, 75% of whom live in urban areas. In 2014, GDP per capita was US \$42,000, making it the fourth largest economy in the world (nominally). Tobacco consumption leads to more than 128,000 deaths each year.

According to the WHO Report on the Global Tobacco Epidemic, 2015, the percentage of current tobacco smokers across both sexes was 24.5% with women smoking at a rate of approximately 20.3%, and men smoking at a rate of 29.0%. In terms of daily users, the rate drops to 20.9% total (17.1% Women and 25.1% Men). For youth aged 12-17, the total smoking rate is 12%; however, unlike adults, young girls have the higher smoking rate over their male counterparts with smoking rates of 12.6% and 11.5% respectively. The use of smokeless forms of tobacco in Germany are very small, with approximately 2% of all adults using smokeless tobacco.

As of December 2014, total government expenditure on tobacco control activities was approximately 4.5 million euros annually.

**Price of Tobacco.** Cigarette prices in Germany are in the middle range of costs across Europe. As of March 2015, the average price per pack of 20 cigarettes was 5.96 euros. Excise taxes on cigarettes meet the recommended percentage of at least 70% excise tax of the retail price set out by the WHO with a 72.9% excise tax in place since 2012.

Smoke-free. As of 2007, Germany passed a comprehensive public smoke-free law. A smoking ban in restaurants, bars, and pubs was brought into force in August 2007, however German courts overturned the ban in one-room bars and restaurants. State authorities may pass more stringent smoke-free laws than those passed by the federal government. As such, regional governments in Bavaria, Saarland, and North Rhine-Westphalia have all introduced stricter smoke-free legislation such as the elimination of designated smoking rooms, or full bans on smoking in public places. Currently smoking is restricted in indoor workplaces and public spaces nationwide. Smoking is also prohibited on all forms of transportation unless 'physically separate units' exist for tobacco users. This means smoking is banned in forms of transportation such as streetcars or trolleys, buses, and taxis.

Tobacco Advertising, Promotion, and Sponsorship. Germany adopted its first advertising and promotion ban of smoked tobacco in 1974 when it passed a comprehensive ban on advertising on both television and radio. A comprehensive advertising ban was later adopted in 1991. Point of sale advertising and promotion is still allowed in Germany. In 2010, a ban on all forms of promotional discounts was passed.

Tobacco Packaging and Labelling. Prior to the European Commission Tobacco Products Directive (TPD), 2014, smoked tobacco products only required one of two text warnings

occupying 30% of the front of the package, as well as an additional text message (one of fourteen authorized messages) on the back of the package occupying 40% of the space. Under the new TPD, Germany must now feature one of 14 combined (graphic) health warnings occupying at least 65% of both the front and back surfaces.

**FCTC Status.** Germany became a party of the FCTC on October 24, 2003 and ratified the Agreement on December 16, 2004.

#### **GREECE**

Greece has an estimated population of 11 million, approximately 78% of whom live in urban areas. As of 2015, GDP per capita was US \$26,000, making it the 46th largest economy in the world (nominally).

According to the WHO Report on the Global Tobacco Epidemic, 2015, the percentage of current tobacco smokers across both sexes was 38.2% with women smoking at a rate of approximately 25.7%, and men smoking at a rate of 51.2%. In terms of daily users, the rate drops to 36.6% total (23.9% Women and 49.7% Men). For youth aged 12-17, the total smoking rate is 16.4% (13.3% female and 19.3% male). The use of smokeless forms of tobacco in Greece is very small, with approximately 0.2% of all adults using smokeless tobacco.

**Price of Tobacco.** Cigarette prices in Greece are low when compared to the rest of Europe. As of March 2015, the average price per pack of 20 cigarettes was 4.36 euros. Excise taxes on cigarettes meet the recommended percentage of at least 70% excise tax of the retail price set out by the WHO with a 79.95% excise tax in place since 2014.

**Smoke-free.** As of July 1, 2009 Greece has banned smoking in all healthcare facilities, food preparation areas, and entertainment venues, as well as public or private working areas, and any enclosed waiting area, airport, or transportation station. While such legislation exists, Greece has not enforced such bans effectively, especially in restaurants, cafes, and bars. As such, few restaurants or cafes comply with the legislation.

**Tobacco Advertising, Promotion, and Sponsorship.** Greece has had a comprehensive ban on all tobacco advertising and promotion since July 2005. As such, all forms of tobacco advertising on television and radio, as well as any domestic print media and outdoor advertising such as billboards are prohibited. Any free distribution of tobacco products is also banned, while promotional discount prices are still allowed.

**Tobacco Packaging and Labelling.** Prior to the European Commission Tobacco Products Directive (TPD), 2014, smoked tobacco products only required text warnings occupying 30% of the primary surface area of the pack. The law required that the back surface of the tobacco package have a warning that covered at least 40% of that surface. Under the new TPD, Greece must now feature one of 14 combined (graphic) health warnings occupying at least 65% of both the front and back surfaces.

FCTC Status. Greece became a party of the FCTC on June 16, 2003 and ratified the Agreement on January 27, 2006.

#### HUNGARY

Hungary has an estimated population of 9.8 million, approximately 71% of whom live in urban areas. As of 2016, GDP per capita was US \$26,941, making it the 58th largest economy in the world (nominally).

According to the latest WHO FCTC Report (2016), the percentage of current tobacco smokers across both sexes was 27.5% with women smoking at a rate of approximately 22.2%, and men smoking at a rate of 33.4%. In terms of daily users, the rate drops to 25.8% total (20.8%) Women and 31.5% Men). For youth aged 13-15, the total smoking rate is 30.5% (28.0% female and 33.0% male).

**Price of Tobacco.** Cigarette prices in Hungary are low when compared to the rest of Europe. As of March 2015, the average price per pack of 20 cigarettes was 3.84 euros. Excise taxes on cigarettes meet the recommended percentage of at least 70% excise tax of the retail price set out by the WHO with a 77.26% excise tax in 2014.

Smoke-free. As of 1999, Hungary has had a comprehensive smoking ban in locations such as: medical institutions, pharmacies, childcare facilities, educational facilities, social institutions, sports facilities, government facilities, hospitality establishments, and workplaces. Under the same law, private establishments could allow smoking under particular circumstances. An amendment to Act XLII of 1999 on the Protection of Non-Smokers and Certain Regulations on the Consumption and Distribution of Tobacco Products was passed by the Hungarian Parliament on 26 April 2011. According to the amendment, by 1 January 2012 smoking is prohibited on all public transportation and in all enclosed public places, including workplaces, bars and restaurants. Smoking is also banned in public education, childcare and health-care institutions; designated areas for smokers will be forbidden both indoors and outdoors at these facilities..

Tobacco Advertising, Promotion, and Sponsorship. Hungary has had a comprehensive ban on all tobacco advertising and promotion since September 2008 (both direct and indirect). Hungary has also banned tobacco company sponsorship in all forms, as well as any use of promotional free-samples of tobacco products. Promotional discounts, as well as advertising at the point-of-sale, are still permitted.

**Tobacco Packaging and Labelling.** Prior to the European Commission Tobacco Products Directive (TPD), 2014, smoked tobacco products required graphic warnings on all tobacco products. Warnings needed to cover 30% of the front and 40% of the back surface areas of all tobacco packages. According to the TPD for 14 text warnings, there are 42 pictures (3 pictures per text). Each year a new picture accompanies the text warnings.

From 20 August 2016, Hungary requires cigarette packages to carry pictorial health warnings of 65% of the front and back of packages. All packs with smaller pictorial warnings will need to be sold out by 20 May 2017.

**FCTC Status.** Hungary became a party of the FCTC on June 16, 2003 and ratified the Agreement on April 7, 2004.

#### **POLAND**

Poland has an estimated population of 38.2 million, approximately 60% of whom live in urban areas. As of 2015, GDP per capita was US \$26,500, and represents the 24th largest economy in the world according to the World Bank.

According to the WHO Report on the Global Tobacco Epidemic, 2015, the percentage of current cigarette smokers across both sexes was 26.0% with women smoking at a rate of approximately 23.0%, and men smoking at a rate of 30.0%. In terms of daily users, the rate drops to 22.0% total (18.0% Women and 27.0% Men). For youth, 12.1% of young females and 15.7% of young males smoke respectively. The use of smokeless forms of tobacco in Poland is very small, with approximately 0.5% of all adults using smokeless tobacco.

**Price of Tobacco.** Cigarette prices in Poland are low when compared to the rest of Europe. As of March 2015, the average price per pack of 20 cigarettes was 3.84 euros. Excise taxes on cigarettes meet the recommended percentage of at least 70% excise tax of the retail price set out by the WHO with a 80.3% excise tax in place as of 2014.

**Smoke-free.** As of April 30, 1996, Poland has had a comprehensive ban on smoking in any premise designated for public use. This includes public transportation and transportation establishments, sporting establishments and public playgrounds for children, workplaces, and public cultural, recreational, food, and entertainment establishments.

**Tobacco Advertising, Promotion, and Sponsorship.** Poland has had a comprehensive ban on all tobacco advertising and promotion since April 30, 1996. As such, all forms of tobacco advertising on television and radio, as well as any domestic print media and outdoor advertising such as billboards are prohibited. This includes a ban on advertising at the point-of-sale, though compliance with this particular area is low according to the WHO. Any form of promotional discount, free-sample, or sponsorship of an event is also banned.

**Tobacco Packaging and Labelling.** Prior to the European Commission Tobacco Products Directive (TPD), 2014, smoked tobacco products only required text warnings occupying 35% of the primary surface area of the pack (30% of the front and 40% of the back). Under the new TPD, Poland must now feature one of 14 combined (graphic) health warnings occupying at least 65% of both the front and back surfaces.

**FCTC Status.** Poland became a party of the FCTC on June 14, 2004 and ratified the Agreement on September 15, 2006.

#### **ROMANIA**

Romania has an estimated population of 21.6 million, approximately 54.6% of whom live in urban areas. As of 2015, GDP per capita was US \$20,800 in Romania, and represents the 51st largest economy in the world according to the World Bank.

According to the WHO Report on the Global Tobacco Epidemic, 2015, the percentage of current cigarette smokers across both sexes was 26.7% with women smoking at a rate of approximately 16.7%, and men smoking at a rate of 37.4%. In terms of daily users, the rate drops to 24.3% total (14.5% Women and 34.9% Men). For youth aged 13-15 the total smoking rate is 11.2%, 10.1% of young females and 12.2% of young males smoking respectively.

**Price of Tobacco.** Cigarette prices in Romania are low when compared to the rest of Europe. As of July 2014, the lowest price per pack of 20 cigarettes was 2.80 euros and the highest price was 3.26 euros inclusive of taxes. Excise taxes on cigarettes meet the recommended percentage of at least 70% excise tax of the retail price set out by the WHO with a 75.4% excise tax in place as of December 2014.

Smoke-free. As of 2002, Romania has had a complete ban on smoking in all enclosed places, including workplaces, public transportation, children's playgrounds, health care facilities, and educational facilities. Smoking is also banned in all restaurants, bars, cafes, and nightclubs.

**Tobacco Advertising, Promotion, and Sponsorship.** Romania has had a comprehensive ban on all tobacco advertising since January 31, 2008. As such, all forms of tobacco advertising on television and radio, as well as print media and outdoor advertising such as billboards are prohibited. Free or paid distribution of tobacco or related products, products that have an evident likeness to tobacco products, and any products used to promote smoking to minors are also banned. As of 2014, promotional discounts on tobacco products were still permitted in Romania.

Tobacco Packaging and Labelling. Graphic health warnings have been required in Romania since 2002. As of 2014, warnings were required to meet a minimum of 35% of the principal display areas (30% on the front and 40% on the back). With the implementation of the European Commission Tobacco Products Directive (TPD), 2014, Romania must now feature one of 14 combined (graphic) health warnings occupying at least 65% of both the front and back surfaces.

FCTC Status. Romania became a party of the FCTC on June 25, 2004 and ratified the Agreement on January 27, 2006.

### **SPAIN**

Spain has an estimated population of 47 million, approximately 79.6% of whom live in urban areas. As of 2015, GDP per capita was US \$28,520 in Spain, and represents the 14th largest economy in the world according to the World Bank.

According to the WHO Report on the Global Tobacco Epidemic, 2015, the percentage of current cigarette smokers across both sexes was 27.0% with women smoking at a rate of approximately 22.8%, and men smoking at a rate of 31.4%. In terms of daily users, the rate drops to 24.0% total (20.2% Women and 27.9% Men). For youth aged 14-18 the total smoking rate is actually higher than that of adults. As of 31 December 2014, the smoking rate among youth was 32.4%, 36.4% of young females and 28.1% of young males smoking respectively.

**Price of Tobacco.** Cigarette prices in Spain are in the middle when compared to the rest of Europe. As of March 2015, the average price per pack of 20 cigarettes was 5.29 euros inclusive of taxes. Excise taxes on cigarettes meet the recommended percentage of at least 70% excise tax of the retail price set out by the WHO with a 78.09% excise tax in place as of 31 July 2014.

Smoke-free. As of January 1, 2006, Spain has had a ban on smoking spaces such as health, teaching, sports, shopping, social, recreational, and entertainment establishments, as well as workplaces, dance halls, gaming, food, and cultural centres. Under this law, smoking rooms are allowed to exist in hospitality establishments (up to 30% of the establishment). All public administrative and law entities are to be smoke free, as are public transportation premises and vehicles, taxis and ambulances. Spain has a strong record of compliance with its smoke-free laws.

Tobacco Advertising, Promotion, and Sponsorship. As of 2003, Spain has banned all advertising from television and radio broadcasting, and all printed mediums (with the exception of tobacco trade publications). Spain has also banned smoking or the mentioning of smoking related brands or activities from all domestic media. Spain has prohibited any promotional activities such as discounts, free distribution, or sponsorships. As of January 2<sup>nd</sup> 2011, the smoke-free legislation was improved with the prohibition of smoking in all hospitality venues with no exceptions as well as at the outdoors of campuses of educational institutions and healthcare centres.

**Tobacco Packaging and Labelling.** Spain mandated graphic health warnings as of May 27, 2010. As of 2014, warnings were required to meet a minimum of 35% of the principal display areas (30% on the front and 40% on the back). With the implementation of the European Commission Tobacco Products Directive (TPD), 2014, Spain must now feature one of 14 combined (graphic) health warnings occupying at least 65% of both the front and back surfaces.

FCTC Status. Spain became a party of the FCTC on June 16, 2003 and ratified the Agreement on January 11, 2005.